CLINICAL TRIAL: NCT03072927
Title: MILD® Percutaneous Image-Guided Lumbar Decompression: A Medicare Claims Study
Status: Recruiting | Type: Observational
Sponsor: Stryker Instruments (Industry)
Responsible Party: Sponsor
Other Study IDs: MILD Medicare Claims
Record Dates: First submitted 2017-02-18; First posted 2017-03-07 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Lumbar Spinal Stenosis
Keywords: Lumbar Spinal Stenosis; Interspinous process decompression; MILD; Medicare; Medicare Advantage
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- MILD: All Medicare patients treated with MILD as reported via CPT® Code 0275T or successor codes (62330/62331).
  Interventions: Device: MILD
- Interspinous Process Decompression: All Medicare patients treated with interspinous process decompression (CPT Code 22869 or 22870, or successor code(s)) for the treatment of LSS with NC.
  Interventions: Device: Interspinous Process Decompression

INTERVENTIONS:
Device: MILD — MILD is performed under fluoroscopic image guidance through an ipsilateral interlaminar dorsal approach to the spine. Partial decompression is performed through the removal of tissue and bone at the symptomatic level confirmed with correlated MRI and clinical findings.
  Groups: MILD
Device: Interspinous Process Decompression — Interspinous Process Decompression
  Groups: Interspinous Process Decompression

SUMMARY:
This prospective longitudinal study will compare incidence rates of Medicare beneficiary surgical and minimally invasive intervention post index procedure, as well as harms associated with the MILD procedure, at 24 months post-treatment with MILD, tested against a control group of similar patients that have had a comparable procedure. This study will start with patients treated with a study procedure having an index date on or after January 1, 2017, and enrollment will continue until stopped by the sponsor.

DETAILED DESCRIPTION:
In this study the treatment group will include all patients receiving MILD, and the control group will include all patients receiving IPD for the treatment of LSS during the enrollment period. Reoperation and harms data will be studied for the MILD and IPD procedures for a 24-month follow-up period after the index procedure using Medicare claims data. This study is exempt from IRB oversight (Department of Health and Human Services regulations 45 CFR 46) and does not require prior enrollment nor patient consent. The inclusion of the study's NCT number on MILD Medicare claims is required and results in enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Medicare beneficiaries receiving MILD or interspinous process decompression
* Diagnosis of LSS with NC

Exclusion Criteria:

* Patients that have received a laminectomy, laminotomy, fusion, interspinous process decompression, or MILD in the lumbar region during the 12 months prior to the index date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study participants will include Medicare beneficiaries for whom claims have been submitted to the Medicare Claims database and who have been enrolled in Medicare fee-for-service or Medicare Advantage for one year prior to their index procedure and two years post index procedure.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2017-03-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of participants with harms associated with the index procedure | 24 months
  Rate of participants with harms associated with the index procedure including, but not limited to, revisions, displacement, mechanical complications, and death. Complications will be counted if they are recorded during the index hospitalization, or any rehospitalization within 30 days of discharge.
Rate of surgical, minimally invasive intervention. | 24 months
  Measure the rate of Medicare beneficiary surgical and minimally invasive intervention for LSS with NC post index procedure.

CONTACTS AND LOCATIONS:
Locations (2168):
- United States (2168):
  - Athens-Limestone Hospital, Athens, Alabama
  - North Baldwin Infirmary, Bay Minette, Alabama
  - Southside Pain Specialists, Birmingham, Alabama
  - St Vincents Birmingham, Birmingham, Alabama
  - The Univ of Alabama At Birmingham, Birmingham, Alabama
  - Birmingham Surgery Center, Birmingham, Alabama
  - Alabama Ortho Spine and Sports, Birmingham, Alabama
  - Outpatient Services East, Birmingham, Alabama
  - St Vincents One Nineteen Health and, Birmingham, Alabama
  - Decatur Ambulatory Surgery Center, Decatur, Alabama
  - Baldwin County Surg Ctr, Fairhope, Alabama
  - Gardendale Surgical Center, Gardendale, Alabama
  - Highland Medical Center, Scottsboro, Alabama
  - Tuscaloosa Surgery Center, Tuscaloosa, Alabama
  - AA Spine & Pain Clinic, Anchorage, Alaska
  - Copper Basin Surg Ctr, Wasilla, Alaska
  - Bullhead City Community Hosp, Bullhead City, Arizona
  - Arizona Specialty Surgery Center, Chandler, Arizona
  - Chandler Surgical Ctr PLC, Chandler, Arizona
  - Advanced Pain Modalities, Chandler, Arizona
  - Northern Arizona Surgicenter, Flagstaff, Arizona
  - Surgery Center at Flagstaff Bone and Joint, Flagstaff, Arizona
  - Mountain View Surgery Center of Gilbert, Gilbert, Arizona
  - Premier Endoscopy Surgery Center, Gilbert, Arizona
  - Santan Surgery Center, Gilbert, Arizona
  - Santa Cruz Valley Regional Hospital, Green Valley, Arizona
  - Havasu Surgery Center, Lake Havasu City, Arizona
  - Banner Surgery Center - Desert, Mesa, Arizona
  - Canyon Surgl Ctr, Mesa, Arizona
  - Mesa Outpatient Treatment Ctr, Mesa, Arizona
  - Rembrandt Outpatient Surgery, Mesa, Arizona
  - Banner Surgery Center - Mesa, Mesa, Arizona
  - Oro Valley Surgical Suites, Oro Valley, Arizona
  - Banner Payson Medical Center, Payson, Arizona
  - Arrowhead North Surgery Center, Peoria, Arizona
  - Banner Surgery Center - Peoria, Peoria, Arizona
  - Palo Verde Pain Specialists ASC, Peoria, Arizona
  - Peoria Foot and Ankle Spclsts, Peoria, Arizona
  - Banner Health Surgicenter, Phoenix, Arizona
  - Banner Surgery Center - Central Phoenix, Phoenix, Arizona
  - Phoenix Eye Surgical Center dba Central Phoenix Surgical Center, Phoenix, Arizona
  - Banner Surg Ctr Biltmore, Phoenix, Arizona
  - Advanced Spine and Pain North Valley, Phoenix, Arizona
  - Optimun Surgical Center, Phoenix, Arizona
  - Arizona Surgical Specialists Center, Phoenix, Arizona
  - JDS Surgical LLC, Phoenix, Arizona
  - Summa Pain Care, Phoenix, Arizona
  - Surgcenter Northern Phoenix LLC, Phoenix, Arizona
  - Prescott OutPatient Surgery Center, Prescott, Arizona
  - Gila Valley Procedure Center, Safford, Arizona
  - South Valley Surgical Center, San Tan Valley, Arizona
  - Arizona Surgl Spclsts Ctr, Scottsdale, Arizona
  - Surgical Centers of Arizona, Scottsdale, Arizona
  - Banner Surg Ctr Desert Vista, Scottsdale, Arizona
  - OrthoArizona Scottsdale Surgery Center, Scottsdale, Arizona
  - Hayden Surgical Center, Scottsdale, Arizona
  - Mountain View Surgery Center of Scottsdale, Scottsdale, Arizona
  - North Valley Surgery Center, Scottsdale, Arizona
  - Virtuous Health Centers III, Scottsdale, Arizona
  - Summit Healthcare Regional Medical Center, Show Low, Arizona
  - Coronado Surgery Center, Sierra Vista, Arizona
  - Banner Sun City West Surgery Center, LLC, Sun City West, Arizona
  - Innovative Surgery Center, Surprise, Arizona
  - Arizona Pain Specialists, LLC, Tempe, Arizona
  - Banner Enticare Tempe Surgery Center, Tempe, Arizona
  - Laser Surgery Center-Tempe, Tempe, Arizona
  - Laser Surgery Center, Tempe, Arizona
  - Pinnacle Outpatient Surgl Instu, Tempe, Arizona
  - Arizona Surgical Specialists Center, Tempe, Arizona
  - Banner Surgery Center, Tucson, Arizona
  - Pain Institute of Southern Arizona Procedure Center, Tucson, Arizona
  - Tucson Med Ctr, Tucson, Arizona
  - Tucson Surgery Center, Tucson, Arizona
  - Banner University Medical Center South, Tucson, Arizona
  - Banner - University Medical Center Tucson, Tucson, Arizona
  - Southern Arizona Va Health Care Sys, Tucson, Arizona
  - Tucson Med Ctr Rincon, Tucson, Arizona
  - Physicians Surgery Center, Blytheville, Arkansas
  - Conway Ambulatory Surgery Center, Conway, Arkansas
  - Fairbanks Memorial Hospital, Fairbanks, Arkansas
  - Northwest Health Physicians' Specialty Hospital, Fayetteville, Arkansas
  - Surgcenter of Fayetteville, Fayetteville, Arkansas
  - Interventional Pain Management Center, Jonesboro, Arkansas
  - Jonesboro Ambulatory Surgery Center, LLC, Jonesboro, Arkansas
  - Outpatient Surgery Center of Jonesboro, Jonesboro, Arkansas
  - NEA Baptist Clinic, Jonesboro, Arkansas
  - VA Medical Center - Little Rock, Little Rock, Arkansas
  - Interventional Surgery Institute, Little Rock, Arkansas
  - Ortho Arkansas, Little Rock, Arkansas
  - Baptist Health Medical Center - Little Rock, Little Rock, Arkansas
  - Central Arkansas Surgery Center, Little Rock, Arkansas
  - Little Rock Surgery Center, Little Rock, Arkansas
  - The Surgical Pavilion, Little Rock, Arkansas
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Executive Surg Ctr of Little Rock, Little Rock, Arkansas
  - Baxter Regional Medical Center, Mountain Home, Arkansas
  - Arkansas Surg Hosp, North Little Rock, Arkansas
  - CVVCA Business, LLC, Pine Bluff, Arkansas
  - Precision Surgical Center of NWA, Rogers, Arkansas
  - Siloam Springs Regional Hospital, Siloam Springs, Arkansas
  - White Hall Ambulatory Surgery Center, White Hall, Arkansas
  - Pacific Ambulatory Surgery Center, Alhambra, California
  - Unicare Surgery Center, Anaheim, California
  - Apple Valley Outpatient Surgical Center, Apple Valley, California
  - St Mary Medical Center, Apple Valley, California
  - SMART Surgery Center, Arcadia, California
  - Sutter Auburn Surgery Center, Auburn, California
  - Delta Bay Surgery Center, LLC, Benicia, California
  - Specialty Surgical Center of Beverly Hills, Beverly Hills, California
  - Surg Ctr of Beverly Hills, Beverly Hills, California
  - Nuvation Pain Group, Buena Park, California
  - On Beach Surgery Center, Buena Park, California
  - Burbank Spine and Pain Surgery Center, Burbank, California
  - Calabasas Surgery Center, Calabasas, California
  - Spanish Hills Surgery Center, Camarillo, California
  - Spine & Sports Surgery Center, Campbell, California
  - Coastal A.S.C, LLC, Carlsbad, California
  - Carlsbad Surgery Center, Carlsbad, California
  - Mercy San Juan Medical Center, Carmichael, California
  - Redwood Surgery Center, Castro Valley, California
  - Golden Springs Surgical Center, Cathedral City, California
  - Chico Surgery Center, Chico, California
  - Enloe Medical Center, Chico, California
  - Deer Creek Surgery Center, Chico, California
  - Surgery Center of California, Chula Vista, California
  - Pain Consultants of San Diego, Chula Vista, California
  - Concourse Diagnostic & Surgical Center, City of Industry, California
  - Am Surg Ctr, Colton, California
  - Premier Outpatient Surgery Center, Colton, California
  - Colusa Med Ctr, Colusa, California
  - Premier Surgery Center, Concord, California
  - Encore Surg Ctr, Covina, California
  - Cmps Surg Ctr, Daly City, California
  - Physicians Surgery Center Of Downey, Downey, California
  - Sutter Elk Grove Surg Ctr, Elk Grove, California
  - Stanford HealthCare Everyville, Emeryville, California
  - Scripps Encinitas Surgery Center, Encinitas, California
  - Specialty Surgl Ctr of Encino, Encino, California
  - Palomar Surgl Ctr, Escondido, California
  - Folsom Surgery Center, Folsom, California
  - Apex Pain and Wellness, Foster City, California
  - Premier Surgery Center, Fountain Valley, California
  - Central Coast Surg Ctr, Freedom, California
  - Palo Alto Med Foundation, Fremont, California
  - Advanced Pain Solutions, Fresno, California
  - Fresno Surgical Hospital, Fresno, California
  - Kaiser Permanente, Fresno, California
  - North Point Surgery Center, Fresno, California
  - Comprehensive Pain Management Center, Fresno, California
  - Herndon Surgery Center, Fresno, California
  - Kaiser Permanente Fresno Medical Center, Fresno, California
  - Renaissance Surgery Center, Fresno, California
  - Summit Surgical, Fresno, California
  - Ky Advanced Surgical Center, Inc., Fresno, California
  - Alliance Surgery Center, Inc, Fullerton, California
  - Laguna Surgery Center, Fullerton, California
  - Avalon Surgery and Robotic Center, Glendale, California
  - Adventist Medical Glendale, Glendale, California
  - Physicians Adventist Surgery Center, Glendale, California
  - Healdsburg District Hospital, Healdsburg, California
  - Hope Ambulatory Surgery Center, Irvine, California
  - Irvine Surgical Partners, LLC, Irvine, California
  - Mission Advanced Pain Mgmt and, Irvine, California
  - Jacobs Med Ctr, La Jolla, California
  - Koman Family Outpatient Pavilion, La Jolla, California
  - Scripps La Jolla Hospital, La Jolla, California
  - EPC Surgery Center, La Mesa, California
  - MemorialCare Surgical Center Laguna Woods, Laguna Woods, California
  - Sutter Lakeside Hospital, Lakeport, California
  - Embassy Surgery Center, Lancaster, California
  - Stanford Hlthcr Tri Valley, Livermore, California
  - Loma Linda University Medical Center, Loma Linda, California
  - VA Medical Center - Loma Linda, Loma Linda, California
  - Lompoc Valley Medical Center, Lompoc, California
  - Shoreline Surgery Center LLC, Long Beach, California
  - Keck Medicine of USC, Los Angeles, California
  - Los Angeles County and Univ of, Los Angeles, California
  - Doctors Outpatient Center for Surgery: DOCS, Los Angeles, California
  - Samaritan Endoscopy Center, Los Gatos, California
  - Silicon Valley ASC, Los Gatos, California
  - Beach Cities Orthopedic Surgery Center, Manhattan Beach, California
  - California Specialty Surgery Center, Mission Viejo, California
  - Minimally Invasive Surgical Institute, Mission Viejo, California
  - Doctors Medical Center Modesto, Modesto, California
  - Modesto Memorial Hospital, Modesto, California
  - Stanislaus Surgical Hospital, Modesto, California
  - Monterey Pain & Spine Institute, Monterey, California
  - Monterey Peninsula Surgery Centers - Munras Ave, Monterey, California
  - Monterey Peninsula Surgery Centers, Monterey, California
  - Mercy Medical Center Mt. Shasta, Mount Shasta, California
  - University Surgery Center, Murrieta, California
  - Loma Linda University Medical Center, Murrieta, California
  - Napa Surgery Center, Napa, California
  - Napa Valley Surgery Center, Napa, California
  - Providence Queen of the Valley Medical Center, Napa, California
  - Newport Coast Surgery Center, Newport Beach, California
  - Regenerative Institute of Newport Beach, Newport Beach, California
  - Heights Surgical Institute, Newport Beach, California
  - Newport Beach Surgery Center, Newport Beach, California
  - North Bay Regional Surgery Center, Novato, California
  - North Coast Surgery Center, Oceanside, California
  - Pacific Surgery Center, Oceanside, California
  - La Veta Surgical Center, Orange, California
  - Oroville Hospital, Oroville, California
  - Stanford Health Care Med Center, Palo Alto, California
  - Stanford Health Care, Palo Alto, California
  - Huntington Ambulatory Surgery Center LLC, Pasadena, California
  - Evolve Restorative Center, Petaluma, California
  - Stanford Health Care ValleyCare, Pleasanton, California
  - Poway Surgery Center, Poway, California
  - Advanced Pain Management, Rancho Mirage, California
  - Rivers Edge Surg Ctr, Rancho Mirage, California
  - Stellar Surgical Specialties, Rancho Mirage, California
  - Apogee Outpatient Surgery Center, Redding, California
  - Court Street Surgery Center, Redding, California
  - Redwood City Medical Center - Kaiser Permanente, Redwood City, California
  - Stanford Health Care, Redwood City, California
  - Kaiser Permanente Richmond Medical Center, Richmond, California
  - Glenwood Surge Ctr, Riverside, California
  - Roseville Surgery Center, Roseville, California
  - Sutter Sierra Surgery Center, Roseville, California
  - Fort Sutter Surgery Center, Sacramento, California
  - Pain Diagnostic and Treatment Center, Sacramento, California
  - UC Davis Medical Cetner-Lawrence Ellison Ambulatory Care Building, Sacramento, California
  - Mercy General Hospital, Sacramento, California
  - Salinas Surgery Center, Salinas, California
  - Natividad Medical Center, Salinas, California
  - San Carlos Clinic, San Carlos, California
  - Scripps Mercy Surgery Pavilion, San Diego, California
  - UCSD Health MOP, San Diego, California
  - Ucsd Med Ctr Hillcrest, San Diego, California
  - UCSD Medical Center, San Diego, California
  - Pacific Surgical Institute, San Diego, California
  - Surgery Center of San Diego, LLC, San Diego, California
  - Rancho Bernardo Surgery Center, San Diego, California
  - VA Medical Center - San Diego, San Diego, California
  - St Lukes Hospital, San Francisco, California
  - San Francisco Hospital, San Francisco, California
  - San Francisco Medical Center, San Francisco, California
  - UCSF Medical Center, San Francisco, California
  - San Gabriel Ambulatory Surgery Center, San Gabriel, California
  - San Gabriel Valley Med Ctr, San Gabriel, California
  - Kaiser Permanente San Jose, San Jose, California
  - Stanford Health Care, San Jose, California
  - Trinity Surgery Center, San Jose, California
  - San Leandro Surgery Center, San Leandro, California
  - Coastal Surgery Center, San Luis Obispo, California
  - Galileo Surgery Center, San Luis Obispo, California
  - Pain Management Specialists, San Luis Obispo, California
  - Hoyman Hong, San Mateo, California
  - San Mateo Surgery Center, San Mateo, California
  - Providence Little Company of Mary Medical Center San Pedro, San Pedro, California
  - Marin Specialty Surgery Center, San Rafael, California
  - UCI Medical Center- Central Distribution Warehouse - Dyer, Santa Ana, California
  - Central Valley Surg Ctr, Santa Barbara, California
  - Coastal Surgery Center, Santa Barbara, California
  - Santa Barbara Outpatient Surgery Center LLC, Santa Barbara, California
  - Palo Alto Med Foundation Warehouse, Santa Clara, California
  - Santa Clarita Surgery Center, Santa Clarita, California
  - Cypress Ambulatory Surgery Center, Santa Maria, California
  - Source Healthcare, Santa Monica, California
  - Source Surgery Center, Santa Monica, California
  - Surgery Center of the Pacific, Santa Monica, California
  - Biohealth Surgl Instu, Santa Monica, California
  - UCLA Medical Center Santa Monica, Santa Monica, California
  - Pacific Restorative Center, Santa Rosa, California
  - Laservue Eye Center, Santa Rosa, California
  - Santa Rosa Surgical Services, Santa Rosa, California
  - St. Joseph Health, Santa Rosa, California
  - Sea Surgery Center, Seal Beach, California
  - Radiance Surgery Center, Sherman Oaks, California
  - Aspen Surgery Center, Simi Valley, California
  - Adventist Health St Helena, St. Helena, California
  - Dameron Hospital, Stockton, California
  - Amb Surg Ctr of Stockton, Stockton, California
  - Stockton Surg Ctr, Stockton, California
  - Ventana Surgical Center, Tarzana, California
  - Innovative Pain Treatment Surgery Center, Temecula, California
  - United Surgery Center-Temecula, Temecula, California
  - Thousand Oaks Surgery Center, Thousand Oaks, California
  - Comprehensive Pain Management Center- St Charles Surgical Center, Thousand Oaks, California
  - Saxon Surgery Center, Thousand Oaks, California
  - St Charles Surgical Center, Thousand Oaks, California
  - UCLA-Thousand Oaks, Thousand Oaks, California
  - Surgery Center of South Bay, Torrance, California
  - Coast Surgery Center of South Bay, Torrance, California
  - Sutter Tracy Community Hospital, Tracy, California
  - David Grant USAF Medical Center, Travis Air Force Base, California
  - Foothill Reg Med Ctr, Tustin, California
  - Ctr For Ortho Surg, Van Nuys, California
  - Desert Valley Hospital, Victorville, California
  - Courtyard Surgery Pavilion, Visalia, California
  - Bass Surgery Center, Walnut Creek, California
  - Queen of the Valley Hosp, West Covina, California
  - Synergy Surgical Center, LLC, Westlake Village, California
  - Orange County Surgery Center, Westminster, California
  - Frank R Howard Mem Hosp, Willits, California
  - Surgery Center of the Rockies, Aurora, Colorado
  - Centeno-Schultz Clinic, Broomfield, Colorado
  - Audubon Surgery Center, Colorado Springs, Colorado
  - Ascent Surg Ctr, Colorado Springs, Colorado
  - ASC at St. Francis, Colorado Springs, Colorado
  - Dry Creek Surgery Center, Englewood, Colorado
  - Englewood Surgery Center, Englewood, Colorado
  - Synergy Surg Ctr, Englewood, Colorado
  - Harmony Surgery Center, Fort Collins, Colorado
  - Family Health West Hospital, Fruita, Colorado
  - Golden Ridge Surgery Center, Golden, Colorado
  - Red Rocks Surgery Center, Golden, Colorado
  - Redlands Mesa Surgery Center, Grand Junction, Colorado
  - Centrum Surgical Center, Greenwood, Colorado
  - Colorado Premier Surgery Center at Greenwood Village, Greenwood Village, Colorado
  - St Anthony Hospital, Lakewood, Colorado
  - Highline South Ambulatory Surgery Center, LLC, Littleton, Colorado
  - Summit View Surgery Center, Littleton, Colorado
  - The Surgery Center at Lone Tree, Lone Tree, Colorado
  - Lincoln Surgery Center, Parker, Colorado
  - Clear Creek Surgery Center, Wheat Ridge, Colorado
  - Surgical Center of Connecticut, Bridgeport, Connecticut
  - HHC Southington Surgery Center, LLC, DBA Cheshire Surgery Center, Cheshire, Connecticut
  - SCA Danbury Surgery Center, Danbury, Connecticut
  - Western Connecticut Orthopedic Surgical Center, Danbury, Connecticut
  - Fairfield Surgery Center, Fairfield, Connecticut
  - Connecticut Surgery Center, Farmington, Connecticut
  - Yale New Haven Health-Greenwich Hospital, Greenwich, Connecticut
  - SCA Guilford Surgery Center, Guilford, Connecticut
  - Hartford Hospital, Hartford, Connecticut
  - Middlesex Hospital, Middletown, Connecticut
  - Yale New Haven Hosp St Raphael Cmps, New Haven, Connecticut
  - Yale New Haven Hosp, New Haven, Connecticut
  - North Haven Surgery Center, North Haven, Connecticut
  - Norwalk Surgery Center, Norwalk, Connecticut
  - Ridgefield Surgical Center, Ridgefield, Connecticut
  - Sasco Hill Surgery Center, Southport, Connecticut
  - The Charlotte Hungerford Hospital, Torrington, Connecticut
  - West Hartford Surgery Center, West Hartford, Connecticut
  - Southwest Connecticut Surgery Center, Wilton, Connecticut
  - Glasgow Surgery Center, Newark, Delaware
  - Delaware Outpatient Center for Surgery, Newark, Delaware
  - Christiana Surgicenter, Newark, Delaware
  - Outpatient Procedure Ctr, Wilmington, Delaware
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - MedStar Health at Lafayette Center, Washington D.C., District of Columbia
  - George Washington Univ Hosp, Washington D.C., District of Columbia
  - Washington Dc Va Med Ctr, Washington D.C., District of Columbia
  - Advanced Asc, Altamonte Springs, Florida
  - AdventHealth Orlando, Apopka, Florida
  - Aventura Hospital and Medical Center, Aventura, Florida
  - Surgery Center of Aventura, Aventura, Florida
  - Boca Raton Surgery Center, Boca Raton, Florida
  - Boca Raton Regional, Boca Raton, Florida
  - Asc of Boca Raton, Boca Raton, Florida
  - Trails Edge Surgery center LLC, Bonita Springs, Florida
  - Boynton Beach Ambulatory Surgery Center, Boynton Beach, Florida
  - Orthopedic Surgery Center of Palm Beach County, Boynton Beach, Florida
  - Specialized Outpatient Surg Ctr For, Boynton Beach, Florida
  - Beth Ambulatory Surgery Center, Boynton Beach, Florida
  - Riverwalk Ambulatory Surgery Center, Bradenton, Florida
  - Musculoskeletal Ambulatory Surgery Center, Bradenton, Florida
  - Musculoskeletal Ambulatory Surgery Centers at Coastal Orthopedics & Sports Medicine, Bradenton, Florida
  - Surgery Center at Pointe West - Lena Rd, Bradenton, Florida
  - Brandon Ambulatory Surgery Center, Brandon, Florida
  - Cape Coral Surg Ctr, Cape Coral, Florida
  - The Ohio Pain Clinic, Centerville, Florida
  - Belleair Surgery Center Ltd, Clearwater, Florida
  - Advanced Surgical Care of Clearwater, Clearwater, Florida
  - South Lake Hosp, Clermont, Florida
  - ParkCreek Surgery Center - Parent, Coconut Creek, Florida
  - ParkCreek Surgery Center, Coconut Creek, Florida
  - Advanced Surgery Center of Coral Gables, Coral Gables, Florida
  - The Gables Surgical Center, Coral Gables, Florida
  - Pohlman Pain Assocs, Coral Springs, Florida
  - Surgery Center at Coral Springs, Coral Springs, Florida
  - Adventhealth Heart Of Florida, Davenport, Florida
  - Davenport Ambulatory Surgery Center, Davenport, Florida
  - Atlantic Surgery Center, Daytona Beach, Florida
  - East Coast Surgery Center, Daytona Beach, Florida
  - Delray Beach Surgery center, Delray Beach, Florida
  - Pohlman Pain Associates, Delray Beach, Florida
  - The Outpatient Center of Delray, Delray Beach, Florida
  - Delray Beach Surgical Suites, Delray Beach, Florida
  - National Pain Institute, Delray Beach, Florida
  - Sacred Heart Med Park at Desitin, Destin, Florida
  - SurgCenter Dunedin, Dunedin, Florida
  - Fort Lauderdale Heart and Rhythm, Fort Lauderdale, Florida
  - Fort Lauderdale Pain Medicine, Fort Lauderdale, Florida
  - Holy Cross Hospital, FTL, Fort Lauderdale, Florida
  - Cypress Creek Outpatient Surgical Center, Fort Lauderdale, Florida
  - Physicians Outpatient Surgery Center, Fort Lauderdale, Florida
  - National Spine and Ortho Surgery Center - Fort Myers, Fort Myers, Florida
  - Gladiolus Surgery Center LLC, Fort Myers, Florida
  - Performance Health Surgery Center, Fort Myers, Florida
  - Advanced Pain Mgmt Spclsts, Fort Myers, Florida
  - Park Center for Procedures, Fort Myers, Florida
  - Colonial Outpatient Surgery Center LLC, Fort Myers, Florida
  - Surg Spclsts Asc, Fort Walton Beach, Florida
  - UF Health Shands Hospital, Gainesville, Florida
  - North Florida Surgical Pavillion, Gainesville, Florida
  - Surgery Center of North Florida, LLC, Gainesville, Florida
  - Orthopaedic Surgery Center, Gainesville, Florida
  - VA Hospital - Gainsville, Gainesville, Florida
  - Hallandale Outpatient Surgical Center, Hallandale, Florida
  - Palmetto Lakes Surgical Center, Hialeah, Florida
  - Hollywood Regional Surgery Center, Hollywood, Florida
  - Memorial Regional Hospital South, Hollywood, Florida
  - Broward Specialty Surgical Center, Hollywood, Florida
  - Univ of Florida Health Jacksonville, Jacksonville, Florida
  - First Coast Surgery Center, Jacksonville, Florida
  - Centurion Surgery Center of Jacksonville, Jacksonville, Florida
  - Mayo Clinic, Jacksonville, Florida
  - River City Surg Ctr, Jacksonville, Florida
  - Riverside Surgical Center, Jacksonville, Florida
  - Touchton Surgery Center, Jacksonville, Florida
  - Point Meadows Surg Ctr, Jacksonville, Florida
  - Surgcenter of Greater Jacksonville, LLC, Jacksonville, Florida
  - Jacksonville Beach Surgery Center, Jacksonville Beach, Florida
  - Advanced Pain Management and Wellness Center, Jupiter, Florida
  - Jupiter Outpatient Surgery Center, Jupiter, Florida
  - National Pain Institute - Lady Lake, Lady Lake, Florida
  - Santa Fe Surgery Center LLC, Lady Lake, Florida
  - Lake City Surg Ctr, Lake City, Florida
  - Lake Mary Surgery Center, Lake Mary, Florida
  - Rinehart Surgery Center, Lake Mary, Florida
  - Lake Worth Surgical Center, Lake Worth, Florida
  - Surgcenter Pinellas, Largo, Florida
  - The Surgery Center of Ft. Lauderdale, Lauderdale Lakes, Florida
  - South Seminole Medical Center, Longwood, Florida
  - Palms West Hospital, Loxahatchee Groves, Florida
  - Palms West Surgicenter, Loxahatchee Groves, Florida
  - Park Place Surgery Center, Maitland, Florida
  - Northwest Medical Center, Margate, Florida
  - Melbourne Surgery Center, Melbourne, Florida
  - Central Florida Spine & Pain, Melbourne, Florida
  - Intracoastal Surgery Center, Melbourne, Florida
  - Merritt Island Surgery Center, Merritt Island, Florida
  - Space Coast Surgery Center, Merritt Island, Florida
  - Coral Gables Surgery Center, Miami, Florida
  - Kw Neurospine, Miami, Florida
  - Coral Gables Hospital, Miami, Florida
  - Univ of Miami Sylvester, Miami, Florida
  - South Miami Hospital, Miami, Florida
  - Northshore Medical Center, Miami, Florida
  - Surgical Park Center, Miami, Florida
  - Surgery Center at Doral, Miami, Florida
  - Miami Surgical Suites LLC, Miami, Florida
  - Miami Surgical Center, Miami, Florida
  - Baptist Hospital of Miami, Miami, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Middleburg Surgery Center, Middleburg, Florida
  - Surgicare of Miramar, Miramar, Florida
  - Mem Hosp Miramar, Miramar, Florida
  - Surgery Center of Mt Dora, Mt. Dora, Florida
  - Surgical Center of Mount Dora, Mt. Dora, Florida
  - Physicians Day Surgery, Naples, Florida
  - Seaside Surgery Center, Naples, Florida
  - Surgery Center of Naples, Naples, Florida
  - North Naples Surgery Center, Naples, Florida
  - Physicians Regional Pine Ridge, Naples, Florida
  - UHealth Miami Med Ctr, North Miami, Florida
  - Coral Ridge Outpatient Center, Oakland Park, Florida
  - Holy Cross Hosp Pain Mgmt, Oakland Park, Florida
  - Advanced Surgl Care of Ocala, Ocala, Florida
  - Central Florida Endoscopy and Surgical Institute of Ocala, Ocala, Florida
  - Marion Surgery Center LLC, Ocala, Florida
  - Ocala Regional Medical Center, Ocala, Florida
  - Orthopedic Institute of Ocala Surgery Center, Ocala, Florida
  - Ocala Surgical Ctr, Ocala, Florida
  - Surgery Center of Ocala, Ocala, Florida
  - West Marion Community Hospital, Ocala, Florida
  - Jacksonville Outpatient Surgery Center, Orange Park, Florida
  - Clay Surgery Center, Orange Park, Florida
  - Downtown Surgery Center, Orlando, Florida
  - AdventHealth Pain Medicine Orlando, Orlando, Florida
  - Jewett Orthopedic Institute Surgery Center, Orlando, Florida
  - Orlando Health Amb Care Ctr, Orlando, Florida
  - Orlando Orthopaedic Outpatient Surgery Center LLC, Orlando, Florida
  - Orlando Regional Medical Center, Orlando, Florida
  - Millenia Surgery Center, Orlando, Florida
  - Orlando Outpatient Surgery Center, Orlando, Florida
  - Alliance Specialty Surgery Center, Ormond Beach, Florida
  - Palm Beach Gardens Regional Surgery Center, Palm Beach, Florida
  - Laser And Surgery Center, Palm Beach Gardens, Florida
  - North County Surgicenter, Palm Beach Gardens, Florida
  - Surgcenter of Palm Beach Gardens, Palm Beach Gardens, Florida
  - Memorial Same Day Surgery Center, Pembroke Pines, Florida
  - Clearway Pain Solutions, Pensacola, Florida
  - West Park Ambulatory Surgery Center, Pinellas Park, Florida
  - Murdock Ambulatory Surgery Center, Port Charlotte, Florida
  - Gulf Pointe Surgery Center, Port Charlotte, Florida
  - Blue Water Surgery Center FL, Port Saint Lucie, Florida
  - St. Lucie Surgery Center, Port Saint Lucie, Florida
  - The Surgical Center of the Treasure Coast, Port Saint Lucie, Florida
  - National Pain Institute, Port Saint Lucie, Florida
  - SurgCenter of St. Lucie, Port Saint Lucie, Florida
  - Sun City Ambulatory Surgery Center, Ruskin, Florida
  - Flagler Surgery Center, Saint Augustine, Florida
  - Orlando Health Medical Pavilion - St. Cloud, Saint Cloud, Florida
  - Orlando Regional St. Cloud, Saint Cloud, Florida
  - Sarasota Surgery Center, Sarasota, Florida
  - Advanced Surgery Center of Sarasota LLC, Sarasota, Florida
  - Premier Surgery Center of Sarasota, Sarasota, Florida
  - Bayview Surgery Center, Sarasota, Florida
  - Florida Pain Management Associates, PA, Sebastian, Florida
  - Sebastian River MC Steward, Sebastian, Florida
  - Bone & Joint Surgical Suites, Sebring, Florida
  - Adventhealth Sebring, Sebring, Florida
  - Larkin Community Hospital, South Miami, Florida
  - Medical Arts Surgery Center at South Miami, South Miami, Florida
  - South Florida Surgery Center, South Miami, Florida
  - Bayfront Health St. Petersburg, St. Petersburg, Florida
  - Florida Physical Medicine, St. Petersburg, Florida
  - Skyway Surgery Center, St. Petersburg, Florida
  - Surgcenter NorthEast, St. Petersburg, Florida
  - Florida Specialty Surgery Center, St. Petersburg, Florida
  - Healthsouth Sunrise Rehab Hospital, Sunrise, Florida
  - Armenia Ambulatory Surgery Center, Tampa, Florida
  - Select Physicians Surgery Center, Tampa, Florida
  - West Florida Surgical Suites, Tampa, Florida
  - South Tampa Surgery Center, LLC, Tampa, Florida
  - Ambulatory Surgery Center, Tampa, Florida
  - Habana Ambulatory Surgery Center, Tampa, Florida
  - Ctr For Advanced Surgical Spclsts, Tampa, Florida
  - The Surgery Center at TGH Brandon Healthplex, Tampa, Florida
  - Westchase Surgery Center, Tampa, Florida
  - Premier Surgical Center, Tavares, Florida
  - Advanced Surg Ctr At Brownwood, The Villages, Florida
  - Titusville Surgery Center, Titusville, Florida
  - Surgery Center at St. Andrews, Venice, Florida
  - Venice Regional Bayfront Health, Venice, Florida
  - Bayfront Venice Reg Surgery, Venice, Florida
  - Sunset Lake Surg Ctr, Venice, Florida
  - Grove Place Surgery Center, Vero Beach, Florida
  - Indian River Medical Center, Vero Beach, Florida
  - The Advanced Center for Surgery, Vero Beach, Florida
  - Vero Beach Surgery Center, Vero Beach, Florida
  - Wellington Endoscopy Center, Wellington, Florida
  - B3 Medical, Wesley Chapel, Florida
  - Surgery Center of Florida, Wesley Chapel, Florida
  - Apollo Surgery Center, West Melbourne, Florida
  - Bethesda Outpatient Surgery Center, West Palm Beach, Florida
  - JFK Medical Center North Campus, West Palm Beach, Florida
  - Northpoint Surgery Center, West Palm Beach, Florida
  - Palm Beach International Surgery Center at The Paley Institute, West Palm Beach, Florida
  - Cleveland Clinic of Weston, Weston, Florida
  - Summerport Surgery Center, Windermere, Florida
  - Day Surg Ctr, Winter Haven, Florida
  - Winter Haven Ambulatory Surgical Center, Winter Haven, Florida
  - National Pain Institute, Winter Park, Florida
  - Florida Hospital Zephyrhills, Zephyrhills, Florida
  - Center for Spine Interventions ASC, LLC (ASC3), Acworth, Georgia
  - Bacon County Hospital, Alma, Georgia
  - Pain Physicians of Atlanta, Alpharetta, Georgia
  - GA Interventional Pain-L, LLC, Athens, Georgia
  - Grady Health System, Atlanta, Georgia
  - Pain Consultants of Atlanta, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - Atlanta Ctr For Ent, Atlanta, Georgia
  - Atlanta Outpatient Surg Ctr, Atlanta, Georgia
  - Alliance Spine and Pain Ctrs, Atlanta, Georgia
  - Peachtree Orthopedics Surgery Center, Atlanta, Georgia
  - Charlie Norwood Va Med Ctr, Augusta, Georgia
  - Summit Spine and Joint Ctr, Augusta, Georgia
  - AOS Surgery Center, Augusta, Georgia
  - Augusta Pain Center, Augusta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - VA Medical Center Augusta, Augusta, Georgia
  - GA Interventional Pain-B, LLC, Braselton, Georgia
  - Premier Surgery Center, Brunswick, Georgia
  - Brunswick Pain Treatment Center, Brunswick, Georgia
  - Alliance Spine and Pain Ctrs, Canton, Georgia
  - GA Interventional Pain-E, LLC, Canton, Georgia
  - Northside Hosp Cherokee, Canton, Georgia
  - Alliance Spine and Pain Ctrs, Carrollton, Georgia
  - GA Interventional Pain-H, LLC, Carrollton, Georgia
  - Tanner Medical Center, Carrollton, Georgia
  - West Georgia Surg Ctr, Carrollton, Georgia
  - Alliance Spine and Pain Ctrs, Cartersville, Georgia
  - Nexus Pain Center, Columbus, Georgia
  - GA Interventional Pain-K, LLC, Conyers, Georgia
  - MD Pain Care, PC, Conyers, Georgia
  - Alliance Covington, Covington, Georgia
  - GA Interventional Pain-C, LLC, Cumming, Georgia
  - Alliance Spine and Pain Ctrs, Dallas, Georgia
  - Ctr For Spine Interventions, Dallas, Georgia
  - GA Interventional Pain-G, LLC, Dalton, Georgia
  - Hamilton Amb Surg Ctr, Dalton, Georgia
  - GA Interventional Pain-D, LLC, Decatur, Georgia
  - Emory Decatur Hosp, Decatur, Georgia
  - Southeastern Orthopaedics Surgery Center, Douglas, Georgia
  - Alliance Spine and Pain Ctrs, Douglasville, Georgia
  - Evans Procedure Center,LLC, Evans, Georgia
  - Pain Consultants of Atlanta, Fayetteville, Georgia
  - Natl Spine and Pain Ctrs, Gainesville, Georgia
  - Northeast Georgia Surgery Center, Gainesville, Georgia
  - Griffin Ctr For Pain and Spine, Griffin, Georgia
  - Southern Pain and Spine - Jasper, Jasper, Georgia
  - Emory Johns Creek, Johns Creek, Georgia
  - Alliance Spine and Pain Ctrs, Lawrenceville, Georgia
  - GA Interventional Pain, LLC, Lawrenceville, Georgia
  - Gwinnett Med Ctr, Lawrenceville, Georgia
  - Revive Ortho Spne and Sports, Lithia Springs, Georgia
  - Athens Orthopedic Clinic (Loganville ASC), Loganville, Georgia
  - Hemlock Ambulatory Surgery Center, Macon, Georgia
  - Alliance Spine and Pain Ctrs, Marietta, Georgia
  - Non Surgical Orthopaedic, Marietta, Georgia
  - Cancer Treatment Ctrs of America At, Newnan, Georgia
  - Georgia Pain and Spine Care, Newnan, Georgia
  - Alliance Spine and Pain, Peachtree City, Georgia
  - GA Interventional Pain-I, LLC, Rome, Georgia
  - GA Interventional Pain- F, LLC, Roswell, Georgia
  - Wellstar North Fulton Hospital, Roswell, Georgia
  - Summit Spine and Joint Ctr Savannah, Savannah, Georgia
  - GA Interventional Pain-J, LLC, Stockbridge, Georgia
  - Pain Care Center of Georgia, Stockbridge, Georgia
  - Alliance Surg Ctr At Johns Creek, Suwanee, Georgia
  - Burke Health Pain Management, Waynesboro, Georgia
  - Samson Pain Center (ASC), Woodstock, Georgia
  - Bingham Memorial Hospital, Blackfoot, Idaho
  - Pain Care Boise, Boise, Idaho
  - Saint Alphonsus Medical Center Boise, Boise, Idaho
  - St. Alphonsus Medical Center (Boise), Boise, Idaho
  - St Lukes Health System, Boise, Idaho
  - North Idaho Pain Center, Coeur d'Alene, Idaho
  - Mountain View Hospital, Idaho Falls, Idaho
  - Idaho Physical Medicine and Rehabilitation, Meridian, Idaho
  - St. Alphonsus Medical Center Nampa, Nampa, Idaho
  - Northwest Specialty Hospital, Post Falls, Idaho
  - Franklin County Hosp, Preston, Idaho
  - Alton Memorial Hospital, Alton, Illinois
  - OSF Saint Anthony Medical Center, Alton, Illinois
  - Associated Surgical Center, Arlington Heights, Illinois
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Northwest Surgicare, Arlington Heights, Illinois
  - Advocate Good Shepard Hospital, Barrington, Illinois
  - Barrington Pain and Spine Institute LLC, Barrington, Illinois
  - Magna Surgical Cente, Bedford Park, Illinois
  - Memorial Hospital Belleville, Belleville, Illinois
  - Swedish American Med Ctr Belvidere, Belvidere, Illinois
  - OSF St. Joseph Medical Center, Bloomington, Illinois
  - Ireland Grove Center for Surgery, Bloomington, Illinois
  - The Center For Outpatient Medicine, Bloomington, Illinois
  - Adventist Bolingbrook Hospital, Bolingbrook, Illinois
  - Oak ASC, LLC, Bourbonnais, Illinois
  - Southern Illinois Healthcare Distribution Center, Carbondale, Illinois
  - Carle Champaign Surgicenter, Champaign, Illinois
  - River North Same Day Surgery, Chicago, Illinois
  - Rush SurgiCenter, Chicago, Illinois
  - Rush Univ Med Ctr, Chicago, Illinois
  - UIC Medical Center- University of Illinois Medical Center, Chicago, Illinois
  - Hyde Park Same Day Surgicenter, LLC, Chicago, Illinois
  - Insight Hospital & Medical Center-Chicago, Chicago, Illinois
  - Swedish Amb Surg Ctr, Chicago, Illinois
  - Swedish Covenant Hosp, Chicago, Illinois
  - University of Chicago Medical Center, Chicago, Illinois
  - Weiss Memorial Hospital, Chicago, Illinois
  - Advanced Ambulatory Surgery Center, Chicago, Illinois
  - Golf Surgical Center, Des Plaines, Illinois
  - Katherine Shaw Bethea Hospital, Dixon, Illinois
  - Good Samaritan Hospital, Downers Grove, Illinois
  - Midwest Center for Day Surgery, Downers Grove, Illinois
  - Pekin Memorial Hospital, East Peoria, Illinois
  - Anderson Surgery Center, Edwardsville, Illinois
  - Effingham Amb Surg Ctr, Effingham, Illinois
  - Advocate Sherman Hospital, Elgin, Illinois
  - Illinois Back and Neck Institute, Elmhurst, Illinois
  - Evanston Hospital Northshore University Health System, Evanston, Illinois
  - North Shore University Evanston Hospital, Evanston, Illinois
  - AMITA St. Francis Hospital, Evanston, Illinois
  - Little Company of Mary Hospital, Evergreen Park, Illinois
  - FHN Memorial Hospital, Freeport, Illinois
  - Gibson Area Hosp and Health Svcs, Gibson City, Illinois
  - Edwardsville Ambulatory Surgery Center LLC, Glen Carbon, Illinois
  - AdventHealth GlenOaks, Glendale Heights, Illinois
  - Adventist Glenoaks Hospital, Glendale Heights, Illinois
  - Herrin Hospital, Herrin, Illinois
  - Highland Park Hospital Northshore University Health System, Highland Park, Illinois
  - AMITA Health Adventist Medical Center Hinsdale, Hinsdale, Illinois
  - Hinsdale Surgical Center, Hinsdale, Illinois
  - AMITA Health St. Alexius Medical Center Hoffman Estates, Hoffman Estates, Illinois
  - Presence St Joseph Med Ctr, Joliet, Illinois
  - Riverside Med Ctr, Kankakee, Illinois
  - Northwestern Lake Forest, Lake Forest, Illinois
  - Advocate Condell Medical Center, Libertyville, Illinois
  - Lindenhurst Surgery Center, Lindenhurst, Illinois
  - Duly Surg Ctr Lombard, Lombard, Illinois
  - Anderson Hospital, Maryville, Illinois
  - Sarah Bush Lincoln Health Ctr, Mattoon, Illinois
  - Centegra Hosp McHenry, McHenry, Illinois
  - Northwestern McHenry Hospital, McHenry, Illinois
  - Center For Minimally Invasive Surgery, Mokena, Illinois
  - Quad City Ambulatory Surgery Center, Moline, Illinois
  - Illinois Sports Medicine & Orthopedic Surgery Center, Morton Grove, Illinois
  - Edward Hospital, Naperville, Illinois
  - Naperville Surgery Center, Naperville, Illinois
  - Silver Cross Surgery Center, New Lenox, Illinois
  - Carle BroMenn Medical Center, Normal, Illinois
  - Oak Brook Surg Ctr, Oak Brook, Illinois
  - Rush Oak Brook Surgery Center, Oak Brook, Illinois
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Rush Oak Park Hospital, Oak Park, Illinois
  - Loyola Ambulatory Surgery Center at Oakbrook, Oakbrook Terrace, Illinois
  - Preferred Surgicenter, Orland Park, Illinois
  - Edgar County Hospital, Paris, Illinois
  - Horizon Health, Paris, Illinois
  - UnityPoint Methodist Comprehensive Pain Management Center, Peoria, Illinois
  - Carle Foundation Hosp, Peoria, Illinois
  - Rochelle Community Hospital, Rochelle, Illinois
  - Swedishamerican Health System, Rockford, Illinois
  - Rockford Ambulatory Surgery Center, Rockford, Illinois
  - OSF Saint Anthony Medical Center, Rockford, Illinois
  - North Pointe Health and Wellness, Roscoe, Illinois
  - Valley Ambulatory Surgery Center, Saint Charles, Illinois
  - Pain Therapy Associates, Schaumburg, Illinois
  - Northshore University Health System, Skokie, Illinois
  - CGH Medical Center, Sterling, Illinois
  - Ingalls Same Day Surgery, Tinley Park, Illinois
  - Tinley Woods Surgery Center, Tinley Park, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Carle Foundation Hosp, Urbana, Illinois
  - OSF Heart of Mary Medical Center, Urbana, Illinois
  - Hawthorn Surgery Center, Vernon Hills, Illinois
  - Monroe County Surgical Center, Waterloo, Illinois
  - Vista Medical Center East, Waukegan, Illinois
  - Northwestern Medicine Central, Winfield, Illinois
  - SurgiCare LLC, Bloomington, Indiana
  - IU Health Beltway Surgery Center, Carmel, Indiana
  - Kentuckiana Medical Center, Clarksville, Indiana
  - Wellspring Pain Solutions, Columbus, Indiana
  - APAC Surgery Center, II, Crown Point, Indiana
  - Pinnacle Hospital, Crown Point, Indiana
  - Franciscan Health Dyer, Dyer, Indiana
  - ASC For Pain Relief, LLC, Evansville, Indiana
  - Indiana Pain Ctrs Evansville, Evansville, Indiana
  - Pain Management Centers of America, Evansville, Indiana
  - Advance Surg Instu of Evansville, Evansville, Indiana
  - Deaconess Main, Evansville, Indiana
  - IU Health Saxony Ambulatory Surgery Center, Fishers, Indiana
  - IU Health Frankort Hospital, Frankfort, Indiana
  - Methodist Hospitals Northlake, Gary, Indiana
  - Goshen Surg Ctr, Goshen, Indiana
  - South Bend Specialty Surgery Center, Granger, Indiana
  - Center for Southside Surgery, LLC, Greenwood, Indiana
  - Interventional Pain Management, Hobart, Indiana
  - Capitol Street Surgery Center, Indianapolis, Indiana
  - IUH University Hospital, Indianapolis, Indiana
  - Senate Street Surgery Center, Indianapolis, Indiana
  - VA Medical Center Indianapolis, Indianapolis, Indiana
  - Community Surgery Center East, Indianapolis, Indiana
  - IU Health East Beltway Surgery Center, Indianapolis, Indiana
  - Franciscan St Francis Health, Indianapolis, Indiana
  - Prime Surg Ctr, Indianapolis, Indiana
  - Eagle Highlands Surgery Center, Indianapolis, Indiana
  - Indiana Univ Health Methodist Med, Indianapolis, Indiana
  - Center for Special Surgery, Indianapolis, Indiana
  - Beltway Surg Ctr, Indianapolis, Indiana
  - IU Health Multi Specialty Surgery Center, Indianapolis, Indiana
  - Advanced Regional Surgery Center, LLC, Jeffersonville, Indiana
  - Kokomo Ambulatory Surgery Center, Kokomo, Indiana
  - Lafayette Pain Care, Kokomo, Indiana
  - Northwest Health - La Porte, La Porte, Indiana
  - Lafayette Pain Care, Lafayette, Indiana
  - Lafayette Surgery Center, Lafayette, Indiana
  - Witham Health Services, Lebanon, Indiana
  - Broadwest Specialty Surgical Center, LLC, Merrillville, Indiana
  - Methodist Hospitals Southlake, Merrillville, Indiana
  - Franciscan Health Michigan City, Michigan City, Indiana
  - Vanguard Medical Group, Michigan City, Indiana
  - Michiana Surgery Center, Mishawaka, Indiana
  - St. Francis Mooresville Surgery Center, Mooresville, Indiana
  - IU Health Ball Outpatient Surgery Center, Muncie, Indiana
  - Interventional Pain Management, LLC, Munster, Indiana
  - Munster Surg Ctr, Munster, Indiana
  - Serenity Surgical, Munster, Indiana
  - The Center for Minimally Invasive Surgery, Munster, Indiana
  - PMC Regional Hospital, New Albany, Indiana
  - Surgical Center of New Albany, New Albany, Indiana
  - Deaconess Gateway, Newburgh, Indiana
  - Gibson General Hospital, Princeton, Indiana
  - Reid Outpatient Surgery & End, Richmond, Indiana
  - South Bend Clinic ASC, South Bend, Indiana
  - Allied Physicians Surg Ctr, South Bend, Indiana
  - Terre Haute Surgical Center, Terre Haute, Indiana
  - Union Hospital, Terre Haute, Indiana
  - Interventional Pain Mgmt, Valparaiso, Indiana
  - Clearview Eye Surgery Center, Vincennes, Indiana
  - Ames Surgery Center, Ames, Iowa
  - Trinity Bettendorf Hosp, Bettendorf, Iowa
  - St Lukes Hosp, Cedar Rapids, Iowa
  - Mercy Cedar Rapids, Cedar Rapids, Iowa
  - Mercy Medical Center - Clinton, Clinton, Iowa
  - West Lakes Surgery Center, Clive, Iowa
  - Jennie Edmundson Memorial Hospital, Council Bluffs, Iowa
  - Genesis Medical Center, Davenport, Iowa
  - Mississippi Valley Surgery Center, Davenport, Iowa
  - Pain Ctrs of Iowa, Davenport, Iowa
  - De Witt Cmnty Hosp, De Witt, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - MercyOne Des Moines Medical Center, Des Moines, Iowa
  - Mason City Surgery Center, Mason City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Dallas County Hospital, Perry, Iowa
  - United Medical Park ASC, LLC, Waterloo, Iowa
  - Allen Memorial Hosp, Waterloo, Iowa
  - UnityPoint Health Waterloo, Waterloo, Iowa
  - Waverly Health Center, Waverly, Iowa
  - Surgery Center of Des Moines West, West Des Moines, Iowa
  - Westown Ambulatory Center, West Des Moines, Iowa
  - St. Lukes Anderson County Hospital, Garnett, Kansas
  - Pain, Spine & Rehab, P.A., Great Bend, Kansas
  - Hays Med Ctr, Hays, Kansas
  - Allen County Hospital, Iola, Kansas
  - Saint Luke's Northland, Kansas City, Kansas
  - Heart of America Surgery, Kansas City, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cushing Memorial Hospital, Leavenworth, Kansas
  - Saint John Hospital, Leavenworth, Kansas
  - Ascentist, Leawood, Kansas
  - Beacon West Surg Ctr, Leawood, Kansas
  - Doctors Hospital, Leawood, Kansas
  - Kansas City Orthopedic Institute, Leawood, Kansas
  - MAO Leawood Surgery Center, LLC, Leawood, Kansas
  - Overland Park Surgery Center, Lenexa, Kansas
  - Advent Health Ottawa, Ottawa, Kansas
  - Menorah Medical Center, Overland Park, Kansas
  - Kansas Surgery Center, Overland Park, Kansas
  - Indian Creek Ambulatory Surgery Center, Overland Park, Kansas
  - South Kansas City Surgicenter, Overland Park, Kansas
  - PainCARE, PA, Overland Park, Kansas
  - Pinnacle Regional Hospital, Overland Park, Kansas
  - Saint Luke's Health System, Overland Park, Kansas
  - Saint Luke's South Surgery Center LLC., Overland Park, Kansas
  - Surgicenter of Johnson County, Overland Park, Kansas
  - Pittsburg Surgical Center, Pittsburg, Kansas
  - Physicians' Surgery Center, Prairie Village, Kansas
  - KU MedWest, Shawnee Mission, Kansas
  - University of Kansas Health System St. Francis Campus, Topeka, Kansas
  - Ascension Via Christi St. Francis, Wichita, Kansas
  - Advanced Pain Medicine Assocs, Wichita, Kansas
  - Kansas Spine & Specialty Hospital, Wichita, Kansas
  - Kansas Surgery & Recovery Center, Wichita, Kansas
  - Kings Daughters Medical Center, Ashland, Kentucky
  - Flaget Memorial Hospital, Bardstown, Kentucky
  - Greenview Surg Ctr, Bowling Green, Kentucky
  - Harrison Memorial Hospital, Cynthiana, Kentucky
  - Central Kentucky Surgery Center, Danville, Kentucky
  - Ephraim McDowell Regional Medical Center, Danville, Kentucky
  - St. Elizabeth - Edgewood, Edgewood, Kentucky
  - St. Elizabeth - Florence, Florence, Kentucky
  - Frankfort Regional Medical Center, Frankfort, Kentucky
  - Owenboro Health Muhlenberg Community Hospital, Greenville, Kentucky
  - Ephraim McDowell James B Haggin Hospital, Hardinsburg, Kentucky
  - Ohio County Hospital, Hartford, Kentucky
  - Deaconess Henderson Hospital, Henderson, Kentucky
  - VA Medical Center - Cooper Dr Div, Lexington, Kentucky
  - Central Baptist Hospital, Lexington, Kentucky
  - The Pain Treatment Center, Inc., Lexington, Kentucky
  - CHI St. Joseph Health Outpatient Surgery Center, Lexington, Kentucky
  - Lexington Clinic Asc, Lexington, Kentucky
  - Lexington Surgery Center, Lexington, Kentucky
  - Saint Joseph Lexington, Lexington, Kentucky
  - UK Interventional Pain Associates, Lexington, Kentucky
  - University Of Kentucky, Lexington, Kentucky
  - Baptist Health Surgery Center, LLC, Lexington, Kentucky
  - Bux Pain Management, Lexington, Kentucky
  - Kentucky Surgery Center, Lexington, Kentucky
  - Paradigm Pain and Spine, Lexington, Kentucky
  - Saint Joseph East Hospital, Lexington, Kentucky
  - Wellward Regenerative Medicine, Lexington, Kentucky
  - Norton Healthcare Inc., Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky
  - Capitol Pain Instu, Louisville, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - Norton St. Matthews, Louisville, Kentucky
  - Norton Audubon Hospital, Louisville, Kentucky
  - Norton Brownsboro Hospital, Louisville, Kentucky
  - Premier Surgery Center of Louisville, Louisville, Kentucky
  - Meadowview Regional Medical Center, Maysville, Kentucky
  - Pikeville Medical Center, Pikeville, Kentucky
  - Clark Regional Medical Center, Winchester, Kentucky
  - Capital Surgical Ctr, Baton Rouge, Louisiana
  - Novamed Surgery Center of Baton Rouge, Baton Rouge, Louisiana
  - Lakeview Reg Med Ctr, Covington, Louisiana
  - Pinnacle Surgery Center, Covington, Louisiana
  - Summit Surg Ctr, Covington, Louisiana
  - Southern Surgical Center, Gray, Louisiana
  - Advanced Pain Institute Treatment Center, Hammond, Louisiana
  - Doctors Outpatient Surgery Center, LLC, Lafayette, Louisiana
  - Lafayette Gen Surgl Hosp, Lafayette, Louisiana
  - Oil Ctr Surgl Plaza, Lafayette, Louisiana
  - Lake Charles Memorial Hospital, Lake Charles, Louisiana
  - Drs Same Day Surg Ctr, Marrero, Louisiana
  - West Jefferson Med Ctr, Marrero, Louisiana
  - Ochsner Clearview Med Complex, Metairie, Louisiana
  - Minden Med Ctr, Minden, Louisiana
  - ArkLaMiss Surgery Center, LLC, Monroe, Louisiana
  - Louisiana Pain Care, Monroe, Louisiana
  - Headache and Pain Ctr, New Iberia, Louisiana
  - Northern Louisiana Medical Center, Ruston, Louisiana
  - Willis-Knighton Medical Center, Shreveport, Louisiana
  - Park Plaza Surgical Specialists, Shreveport, Louisiana
  - Sterling Surgical Hospital, Slidell, Louisiana
  - Thibodaux Regional Health System, Thibodaux, Louisiana
  - Northern Light Eastern Maine Medical Center, Bangor, Maine
  - Northern Light Interventional Pain Management, Bangor, Maine
  - Calais Regional Hospital, Calais, Maine
  - Franklin Memorial Hospital, Farmington, Maine
  - York Hosp, York Village, Maine
  - Clearway Pain Solutions, Annapolis, Maryland
  - Medstar Surg Ctr At Annapolis, Annapolis, Maryland
  - Riva Road Surgery Center, Annapolis, Maryland
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - Johns Hopkins Bayview Medical Center, Baltimore, Maryland
  - MedStar Harbor Hospital, Baltimore, Maryland
  - MedStar Health Harbor Hospital, Baltimore, Maryland
  - Clearway Pain Solutions, Baltimore, Maryland
  - Johns Hopkins Enterprise, Baltimore, Maryland
  - MedStar Franklin Square Medical Center, Baltimore, Maryland
  - MedStar Good Samaritan Hospital, Baltimore, Maryland
  - National Spine and Pain Centers, Bel Air, Maryland
  - Clearway Pain Solutions - Bel Air, Bel Air, Maryland
  - Atlantic General Hospital, Berlin, Maryland
  - Berlin Interventional Pain Management, Berlin, Maryland
  - National Spine and Pain Centers, Berwyn Heights, Maryland
  - Capitol Surgical Center, Bethesda, Maryland
  - Clearway Pain Solutions - Bethesda, Bethesda, Maryland
  - District Surg Ctr, Bethesda, Maryland
  - Johns Hopkins Health Care & Surgery Center - Bethesda, Bethesda, Maryland
  - Surgcenter of the Potomac, Bethesda, Maryland
  - Surgical Specialty Center of Mid-Atlantic, LLC, Bethesda, Maryland
  - Walter Reed Medical Center, Bethesda, Maryland
  - National Spine and Pain Centers, Bowie, Maryland
  - MedStar Southern Maryland Hospital Center, Clinton, Maryland
  - Johns Hopkins Howard County Operating Room, Columbia, Maryland
  - Johns Hopkins Surgery Centr- Howard County, Columbia, Maryland
  - Clearway Pain Solutions - Columbia, Columbia, Maryland
  - National Spine and Pain Centers, Columbia, Maryland
  - Univ of Maryland Orthopaedics, Columbia, Maryland
  - National Spine and Pain Centers, Cumberland, Maryland
  - Clearway Pain Solutions, Dundalk, Maryland
  - Clearway Pain Solutions - Easton, Easton, Maryland
  - Elkridge Ambulatory Surgery Center, Elkridge, Maryland
  - Upper Bay Surgery Center, Elkton, Maryland
  - Ellicott City Ambulatory Surgery Center, Ellicott City, Maryland
  - Monocacy Surgery Center, LLC, Frederick, Maryland
  - National Pain and Spine Centers, Frederick, Maryland
  - Thomas Johnson Surgery Center, Frederick, Maryland
  - National Spine and Pain Centers, Germantown, Maryland
  - Chesapeake Urology Holy Cross, Germantown, Maryland
  - Clearway Pain Solutions, Germantown, Maryland
  - Clearway Pain Solutions, Glen Burnie, Maryland
  - National Spine and Pain Centers, Glen Burnie, Maryland
  - SurgCenter of Glen Burnie, Glen Burnie, Maryland
  - Synergy Spine and Pain Ctr, Glenn Dale, Maryland
  - Hanover Parkway Surgery Center, Greenbelt, Maryland
  - National Spine and Pain Centers, Hagerstown, Maryland
  - Parkway Surgery Center, Hagerstown, Maryland
  - Sports and Spine Pain Management, Havre de Grace, Maryland
  - SurgCenter of Northern Baltimore, LLC, Hunt Valley, Maryland
  - Charles Regional Surgery Center, La Plata, Maryland
  - Advanced Surgical Care of Maryland, Lanham, Maryland
  - Park Center Surgical Center, Laurel, Maryland
  - Precision Ortho and Sports, Laurel, Maryland
  - Leonardtown Surg Ctr, Leonardtown, Maryland
  - MedStar St. Mary's Hospital, Leonardtown, Maryland
  - St Marys Hosp, Leonardtown, Maryland
  - Maryland Specialty Surgery Center, Linthicum Heights, Maryland
  - Johns Hopkins Surg Ctrs Series, Lutherville-Timonium, Maryland
  - Simcare ASC, Mount Airy, Maryland
  - Clearway Pain Solutions - White Marsh, Nottingham, Maryland
  - Johns Hopkins Surgery Center- White Marsh, Nottingham, Maryland
  - Medstar Montgomery Medical Center, Olney, Maryland
  - ClearWay Pain Solutions, Owings Mills, Maryland
  - Clearway Pain Solutions, Owings Mills, Maryland
  - SurgiCenter of Baltimore, Owings Mills, Maryland
  - Adventist Hlthcr Surg Ctr At Natl, Oxon Hill, Maryland
  - Harbor Heights Surg Ctr, Oxon Hill, Maryland
  - Harborside Surg Ctr, Oxon Hill, Maryland
  - National Spine and Pain Centers, Oxon Hill, Maryland
  - Anne Arundel Med Ctr Pavsadena, Pasadena, Maryland
  - National Spine and Pain Centers, Pikesville, Maryland
  - Sapna Surg Ctr of Potomac, Potomac, Maryland
  - Clearway Surgery Center - Prince Frederick, Prince Frederick, Maryland
  - Prince Frederick Surg Ctr, Prince Frederick, Maryland
  - Pain Management Specialists, Rockville, Maryland
  - National Spine and Pain Centers, Rockville, Maryland
  - MedStar Franklin Square Medical Center, Rosedale, Maryland
  - National Spine and Pain Centers, Rosedale, Maryland
  - Peninsula Ortho Assocs Surg Ctr, Salisbury, Maryland
  - Clearway Pain Solutions - Salisbury, Salisbury, Maryland
  - Holy Cross Hospital, Silver Spring, Maryland
  - Clearway Pain Solutions, Stevensville, Maryland
  - Timonium Surgery Center, Timonium, Maryland
  - Ruxton Surgi Center, Towson, Maryland
  - Clearway Pain Solutions Largo, Upper Marlboro, Maryland
  - Largo Medical Center, Upper Marlboro, Maryland
  - ClearWay Pain Solutions, Waldorf, Maryland
  - Clearway Surgery Center - WALDORF ASC, Waldorf, Maryland
  - National Spine and Pain Centers, Waldorf, Maryland
  - Clearway Pain Solutions - Westminster, Westminster, Maryland
  - National Spine and Pain Centers, White Plains, Maryland
  - Saint Anne's Hospital: Southern New England Surgical Center, Attleboro, Massachusetts
  - Sturdy Memorial Hospital, Attleboro, Massachusetts
  - New England Surgery Center, Beverly, Massachusetts
  - Tufts Med Ctr, Boston, Massachusetts
  - Massachusetts Gen Hosp, Boston, Massachusetts
  - Brigham & Womens Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - New England Baptist Hospital, Boston, Massachusetts
  - Brigham and Women's Faulkner Hospital, Boston, Massachusetts
  - St Elizabeth's Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Lahey Clinic Burlington, Burlington, Massachusetts
  - New England Ambulatory SurgiCenter, Cambridge, Massachusetts
  - Lahey Outpatient Center - Danvers, Danvers, Massachusetts
  - Brigham and Women's Foxborough, Foxborough, Massachusetts
  - Brigham and Women's-Mass General Health Care Center, Foxborough, Massachusetts
  - Complete Spine and Pain Care, Framingham, Massachusetts
  - Metrowest Medical Center - Framingham Union Hospital, Framingham, Massachusetts
  - Baystate Medical Center - Holyoke, Holyoke, Massachusetts
  - Holyoke Medical Center Inc, Holyoke, Massachusetts
  - Medford Surg Ctr, Medford, Massachusetts
  - Natick Surg Ctr, Natick, Massachusetts
  - Beth Israel Deaconess Hospital, Needham, Massachusetts
  - Newton Wellesley Hospital Ambulatory Care Center, Newton, Massachusetts
  - New England Pain Care Pain and Wellness Center, Peabody, Massachusetts
  - Berkshire Medical Center, Pittsfield, Massachusetts
  - Beth Israel Deaconess - Plymouth, Plymouth, Massachusetts
  - Salem Hospital, Salem, Massachusetts
  - The Surgery Center, Shrewsbury, Massachusetts
  - Surgery Center of New England, Springfield, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - Baystate Pain Management Center, Springfield, Massachusetts
  - Northeast Ambulatory Center, Stoneham, Massachusetts
  - Morton Hospital, Taunton, Massachusetts
  - Ann Arbor Surgl Ctr, Ann Arbor, Michigan
  - Univ of Michigan Univ Hosp, Ann Arbor, Michigan
  - West Michigan Surgery Center, Big Rapids, Michigan
  - Bloomfield Hills Surgical Center, Bloomfield Hills, Michigan
  - U of M Sparrow Eaton Hospital, Charlotte, Michigan
  - Michigan Neurology Associates & P.C., Clinton Township, Michigan
  - Premier Surgical Center of Michigan, Clinton Township, Michigan
  - Insight Hosp and Med Ctr Coldwater, Coldwater, Michigan
  - Huron Valley Sinai Hospital, Commerce, Michigan
  - Dearborn Surgery Center, Dearborn, Michigan
  - Advanced Surgery Center, Dearborn, Michigan
  - Executive Ambulatory Surgical Center, Dearborn, Michigan
  - Henry Ford Health System - Dearborn, Dearborn, Michigan
  - Associated Surgical Center of Dearborn, Dearborn Heights, Michigan
  - Detroit Receiving Hospital, Detroit, Michigan
  - Rehabilitation Institute of Michigan Main Campus, Detroit, Michigan
  - Rehabilitation Institute of Michigan, Detroit, Michigan
  - Ascension St John Hospital - Detroit, Detroit, Michigan
  - St. John Hospital and Medical Center, Detroit, Michigan
  - Eaton Rapids Med Ctr, Eaton Rapids, Michigan
  - Insight Pain Management - Flint, Flint, Michigan
  - Surgery Center Health Park, Grand Blanc, Michigan
  - Spectrum Health Grand Rapids, Grand Rapids, Michigan
  - Grand Valley Surgical Center, Grand Rapids, Michigan
  - Grand Rapids Surgical Suites, Grand Rapids, Michigan
  - Lake Drive Surgical Center, Grand Rapids, Michigan
  - Michigan Institute for Advanced Surgery, Lake Orion, Michigan
  - Genesis Surgery Center, Lansing, Michigan
  - McLaren Hospital - Lapeer, Lapeer, Michigan
  - Enhance Center for Interventional Spine and Sports, Livonia, Michigan
  - Ascension St. John Hospital Health Center at 23 Mile, Macomb, Michigan
  - Aspire Rural Health System Marlette, Marlette, Michigan
  - Upper Peninsula Surgery Center, Marquette, Michigan
  - Mymichigan Med Ctr Midland, Midland, Michigan
  - Surgical Institute of Monroe, Monroe, Michigan
  - Novi Surgery Center, Novi, Michigan
  - Henry Ford Health System - Columbus, Novi, Michigan
  - Michigan Outpatient Surgical Solutions, Novi, Michigan
  - Memorial Healthcare, Owosso, Michigan
  - Henry Ford Health System- Plymouth, Plymouth, Michigan
  - Blue Water Surgery Center, Port Huron, Michigan
  - Surg Ctr of Kalamazoo, Portage, Michigan
  - Barclay Surg Ctr, Rochester Hills, Michigan
  - Millman-Derr Surgicenter, Rochester Hills, Michigan
  - Kumar Surgical Center, Rochester Hills, Michigan
  - Oakland Surgi Center, Inc., Rochester Hills, Michigan
  - Henry Ford Health System - Royal Oak, Royal Oak, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - Royal Oak Surgical Center, Royal Oak, Michigan
  - Matrix Surgery Center, Saginaw, Michigan
  - Towne Centre Surgery Center, Saginaw, Michigan
  - Sheridan Community Hospital, Sheridan, Michigan
  - Great Lakes Surgical Center, Southfield, Michigan
  - Surgeons Choice Medical Center, Southfield, Michigan
  - Pioneer Endo and Surg Ctr, Sterling Heights, Michigan
  - Three Rivers Health, Three Rivers, Michigan
  - Copper Ridge Surgery Center, Traverse City, Michigan
  - Summit Surgery Center, Troy, Michigan
  - Michigan Advanced Surgical Center, PLLC, Warren, Michigan
  - Southeast Michigan Surgical Hospital, Warren, Michigan
  - Synergy Spine & Orthopedic Surgery Center, LLC, Warren, Michigan
  - American Surgical Centers, West Bloomfield, Michigan
  - MidMichigan Medical Center - West Branch, West Branch, Michigan
  - Genesys Surgery Center LLC, Westland, Michigan
  - Forest Health Medical Center, Ypsilanti, Michigan
  - West Michigan Surgical Center, Zeeland, Michigan
  - Center for Pain Management Ambulatory Surgery, LLC, Alexandria, Minnesota
  - Ctr For Pain Mgmt, Bemidji, Minnesota
  - Sanford Bemidji Med Ctr, Bemidji, Minnesota
  - Twin Cities Pain Clinic- Burnsville, Burnsville, Minnesota
  - Pain Centers of Minnesota, Chaska, Minnesota
  - Two Twelve Surgery Center, Chaska, Minnesota
  - Riverview Health, Crookston, Minnesota
  - Deer River Hlthcare Ctr, Deer River, Minnesota
  - Lakewalk Surgery Center, Duluth, Minnesota
  - Essentia Health - Duluth, Duluth, Minnesota
  - Twin Cities Pain Clinic and Surgery Center, Edina, Minnesota
  - Mankato Clinic Ltd, Mankato, Minnesota
  - Mayo Clinic Health System In, Mankato, Minnesota
  - Twin Cities Surg Ctr Maplewood, Maplewood, Minnesota
  - Nura Precision Pain Management - Edina Clinic, Minneapolis, Minnesota
  - Fairview UMN Health, Minneapolis, Minnesota
  - CentraCare Health Monticello, Monticello, Minnesota
  - Mille Lacs Hosp, Onamia, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - CentraCare Plaza, Saint Cloud, Minnesota
  - St Cloud Hosp, Saint Cloud, Minnesota
  - Center for Pain Management Ambulatory Surgery Center-Sartell, Sartell, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Carris Health Rice Mem Hosp, Willmar, Minnesota
  - CentraCare - Willmar Surgery Center, Willmar, Minnesota
  - RAYUS Radiology - Woodbury ASC, Woodbury, Minnesota
  - Ochsner Med Ctr Hancock, Bay Saint Louis, Mississippi
  - Kings Daughters Med Ctr, Brookhaven, Mississippi
  - Flowood Surgery Center, LLC, Flowood, Mississippi
  - Madison Spine Surg Ctr, Flowood, Mississippi
  - Mississippi Sports Medicine and Ort, Flowood, Mississippi
  - Singing River Gulfport, Gulfport, Mississippi
  - Southern Surgery Center, Hattiesburg, Mississippi
  - Hattiesburg Clinic, Hattiesburg, Mississippi
  - Univ of Mississippi Med Ctr, Jackson, Mississippi
  - Surgicare of Jackson, Jackson, Mississippi
  - South Central Regional Medical Center, Laurel, Mississippi
  - Anderson Regional Health System, Meridian, Mississippi
  - Anderson Regional Medical Center, South Campus, Meridian, Mississippi
  - Anderson Regional Medical Center, Meridian, Mississippi
  - The Pain Management Center of Meridian, Meridian, Mississippi
  - Total Pain Care, Meridian, Mississippi
  - Pain Consultants ASC, Pascagoula, Mississippi
  - Mid South Pain Treatment, Southaven, Mississippi
  - OCH Regional Medical Center, Starkville, Mississippi
  - SOG Surgery Center, Tupelo, Mississippi
  - Vicksburg Spine Ctr, Vicksburg, Mississippi
  - Baptist Med Ctr Yazoo, Yazoo City, Mississippi
  - Harrison County Community Hospital, Bethany, Missouri
  - Citizens Memorial Hospital, Bolivar, Missouri
  - Southeast Hospital, Cape Girardeau, Missouri
  - Auburn Surgery Center, Cape Girardeau, Missouri
  - West Park Surgery Center, Cape Girardeau, Missouri
  - Carroll County Memorial Hospital, Carrollton, Missouri
  - Mercy Hospital Carthage, Carthage, Missouri
  - Interventional Pain Center of Chesterfield, Chesterfield, Missouri
  - Interventional Pain Center Chesterfield - Satellite, Chesterfield, Missouri
  - Hedrick Medical Center, Chillicothe, Missouri
  - NMSC of St. Peters, City of Saint Peters, Missouri
  - St Peters Ambulatory Surgery Center, City of Saint Peters, Missouri
  - Noble Pain Management, Columbia, Missouri
  - Noble Pain Mangement, Columbia, Missouri
  - The Surgery Center of Columbia, Columbia, Missouri
  - The Surgical Center at Columbia Orthopaedic Group, Columbia, Missouri
  - Midamerica Spine Ctr, Creve Coeur, Missouri
  - North Campus Surgery Center, Creve Coeur, Missouri
  - Manchester Surgery Center, Des Peres, Missouri
  - Parkland Health Ctr Farmington, Farmington, Missouri
  - SSM St. Clare Surgical Center, Fenton, Missouri
  - Twin Cities Surgery Center, Festus, Missouri
  - Frontenac Surgery and Spine Center, Frontenac, Missouri
  - SSM Health St. Mary's Hospital - Jefferson City, Jefferson City, Missouri
  - Truman Medical Center, Kansas City, Missouri
  - Briarcliff Surgery Center, Kansas City, Missouri
  - North Kansas City Hospital, Kansas City, Missouri
  - Saint Luke's Hospital Of Kansas City, Kansas City, Missouri
  - Saint Luke's Pain Management Center, Kansas City, Missouri
  - VA Medical Center Kansas City, Kansas City, Missouri
  - Mercy Hosp Lebanon, Lebanon, Missouri
  - Lees Summit Medical Center, Lee's Summit, Missouri
  - Beacon Surgery Center, Lee's Summit, Missouri
  - Midwest Pain Management Center, Lee's Summit, Missouri
  - Liberty Hospital, Liberty, Missouri
  - Fitzgibbon Memorial Hospital, Marshall, Missouri
  - Progress West Hospital, O'Fallon, Missouri
  - Phelps County Regional Medical Center, Rolla, Missouri
  - St Johns Health System Inc, Springfield, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - Ssm Health St Louis Univ Hosp South, St Louis, Missouri
  - Barnes Jewish Hospital - North, St Louis, Missouri
  - Barnes Jewish N Hospital, St Louis, Missouri
  - Barnes Jewish Hospital South, St Louis, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - MidAmerica Spine Center, St Louis, Missouri
  - Advanced Surgical Center of Sunset Hills, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Christian Hospital, St Louis, Missouri
  - Barnes-Jewish West County Hospital, St Louis, Missouri
  - Mercy Hospital of St Louis, St Louis, Missouri
  - Mercy Hospital Lincoln, Troy, Missouri
  - Mercy Hospital Washington, Washington, Missouri
  - West Plains Surgery Center, West Plains, Missouri
  - Bozeman Outpatient Surgery Center, Bozeman, Montana
  - Freeman Health System, Joplin, Montana
  - Bellevue Medical Center, Bellevue, Nebraska
  - Butler County Health Care Center, David City, Nebraska
  - Community Medical Center, Falls City, Nebraska
  - CHI Health St. Francis, Grand Island, Nebraska
  - Grand Island Regional Medical Center, Grand Island, Nebraska
  - Grand Island Surgery Center, Grand Island, Nebraska
  - Heartland Radiology, Grand Island, Nebraska
  - Total Body Pain Institute, Grand Island, Nebraska
  - Thayer County Health Services, Hebron, Nebraska
  - Kearney Pain Treatment Center, Kearney, Nebraska
  - Southwest Lincoln Surgery Center, Lincoln, Nebraska
  - Doctors Outpatient Surgery Center, Lincoln, Nebraska
  - NPI Surgery Center LLC, Lincoln, Nebraska
  - NPI Surgery Center, Lincoln, Nebraska
  - Nebraska Pain Institute, Lincoln, Nebraska
  - Kearney County Health Services, Minden, Nebraska
  - Faith Regional Health Services, Norfolk, Nebraska
  - Faith Regional Surgery Center, Norfolk, Nebraska
  - Fountain Point Surgery Center, Norfolk, Nebraska
  - Advanced Surgery Center, Omaha, Nebraska
  - Nebraska Medical Center, Omaha, Nebraska
  - Meth Hosp, Omaha, Nebraska
  - Omaha Ambulatory Surgery Center, Omaha, Nebraska
  - Pacific Surg Ctr, Omaha, Nebraska
  - Methodist HealthWest, Omaha, Nebraska
  - Village Pointe Health Center, Omaha, Nebraska
  - Lakeside Surgery Center, Omaha, Nebraska
  - Orthonebraska Hosp, Omaha, Nebraska
  - Miracle Hills Surgery Center, Omaha, Nebraska
  - Howard County Medical Center, Saint Paul, Nebraska
  - Regional West Medical Center, Scottsbluff, Nebraska
  - Scottsbluff Surg Ctr, Scottsbluff, Nebraska
  - Brodstone Memorial Hospital, Superior, Nebraska
  - Saunders Medical Center, Wahoo, Nebraska
  - Carson Tahoe Regional Healthcare, Carson City, Nevada
  - Carson Tahoe Regional Medical Center, Carson City, Nevada
  - Sierra Surgery Hospital, Carson City, Nevada
  - William Bee Ririe Hospital, Ely, Nevada
  - VA Medical Center Pecos MSPV, Las Vegas, Nevada
  - Nevada Surgical Suites - Central Location, Las Vegas, Nevada
  - Sahara Surgery Center, Las Vegas, Nevada
  - Red Rock Surgery Center, Las Vegas, Nevada
  - Surgical Arts Center, Las Vegas, Nevada
  - Nevada Surgical Suites, Las Vegas, Nevada
  - Smoke Ranch Surgery Center, Las Vegas, Nevada
  - Speciality Surg Ctr, Las Vegas, Nevada
  - DLJT Management Services, LLC, Las Vegas, Nevada
  - Surgery Center of Reno, Reno, Nevada
  - Quail Surgical and Pain Management Center, Reno, Nevada
  - Nevada Advanced Pain Spclsts, Reno, Nevada
  - Renown South Meadows Medical Center, Reno, Nevada
  - Northern Nevada Medical Center, Sparks, Nevada
  - Humboldt General Hospital, Winnemucca, Nevada
  - Minimally Invasive Surgery Center of New England, Bedford, New Hampshire
  - Wentworth-Douglass Hospital, Dover, New Hampshire
  - Catholic Medical Center, Manchester, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Centers For Pain Solutions, Nashua, New Hampshire
  - New England Center for Orthopaedic Surgery, Portsmouth, New Hampshire
  - Portsmouth Regional Ambulatory Surgery Center, Portsmouth, New Hampshire
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Stratham Ambulatory Surgery Center, Stratham, New Hampshire
  - 877-446-6724, Bayonne, New Jersey
  - Bayonne Medical Center, Bayonne, New Jersey
  - Bloomfield Surgi-Center, Bloomfield, New Jersey
  - Freedom Surgical Center, LLC, Bloomfield, New Jersey
  - Jasper Ambulatory Surgical Center, Brick, New Jersey
  - Seashore Surgical Institute, Brick, New Jersey
  - Performance Surgical Associates, Bridgewater, New Jersey
  - Trinity Surgical and Pain Management dba Performance Surgical Associates, Bridgewater, New Jersey
  - Ambulatory Surgical Center of Somerset, Bridgewater, New Jersey
  - Bridgewater Ambulatory Surgery Center, Bridgewater, New Jersey
  - Cape Regional Medical Center, Cape May Court House, New Jersey
  - Jefferson Surgery Center-Cherry Hill, Cherry Hill, New Jersey
  - Millennium Surgical Center, Cherry Hill, New Jersey
  - Clifton Surgery Center, Inc, Clifton, New Jersey
  - Same Day Procedures, Clifton, New Jersey
  - East Brunswick Surgery Center, East Brunswick, New Jersey
  - RWJ Endosurgical Center, East Brunswick, New Jersey
  - East Orange Gen Hosp, East Orange, New Jersey
  - Camis, Llc, Eatontown, New Jersey
  - Central Jersey Surgery Center, LLC, Eatontown, New Jersey
  - Ambulatory Surgical Center of New Jersey, LLC, Edison, New Jersey
  - Edison Surgery Center, LLC, Edison, New Jersey
  - Menlo Park Surgery Center, Edison, New Jersey
  - Access Surgery Center, Egg Harbor, New Jersey
  - Trinitas Hospital, Elizabeth, New Jersey
  - Inspira Medical Center Elmer, Elmer, New Jersey
  - Health East ASC, Englewood, New Jersey
  - Patient Care Associates, Englewood, New Jersey
  - Englewood Cliffs Surg Ctr, Englewood Cliffs, New Jersey
  - Hunterdon Center for Surgery, Flemington, New Jersey
  - Hunterdon Medical Center, Flemington, New Jersey
  - Hanover Hills Surgery Center LLC, Florham Park, New Jersey
  - Hudson Crossing Surgery Center, Fort Lee, New Jersey
  - SurgiCare of Freehold, LLC, Freehold, New Jersey
  - Hackensack Musculoskeletal Surg Ctr, Hackensack, New Jersey
  - Hackensack Surgery Center, LLC, Hackensack, New Jersey
  - Burlington Asc, Hainesport, New Jersey
  - North American Spine & Pain, Hainesport, New Jersey
  - Hamilton Surgery Center, Hamilton, New Jersey
  - Ambulatory Surgical Pavilion of New Jersey, Hammonton, New Jersey
  - Harrison Endo Surgical Center, Harrison, New Jersey
  - Hoboken Univ Med Ctr, Hoboken, New Jersey
  - Bayshore Hospital, Holmdel, New Jersey
  - Jackson Surgical Center, Jackson, New Jersey
  - Jersey City Medical Center, Jersey City, New Jersey
  - Amb Pain and Disability Mgmt Ctr, Jersey City, New Jersey
  - SurgiCore Jersey City, Jersey City, New Jersey
  - SurgiCore Jersey City, Kenilworth, New Jersey
  - NorthEast Surgicare, LLC, Lakewood, New Jersey
  - Lakewood Surgery Center, Lakewood, New Jersey
  - Reclaimability Pain Svcs, Linwood, New Jersey
  - Parkway Ambulatory Surgery Center, Lyndhurst, New Jersey
  - Manalapan Surgery Center, Manalapan, New Jersey
  - Northern Monmouth Regional Surgery Center, Manalapan, New Jersey
  - Premier Surgical Center, Marlton, New Jersey
  - Vantage Surgery Center, Medford, New Jersey
  - Specialty Surgery Center of Middletown, Middletown, New Jersey
  - SurgiCore Rockland and Bergen Surgery Center, Montvale, New Jersey
  - Morristown Memorial Pain Mgmt, Morristown, New Jersey
  - Memorial Ambulatory Surgery Center LLC, Mount Holly, New Jersey
  - Fellowship Surgery Center, Mount Laurel, New Jersey
  - Surgical Center of South Jersey, Mount Laurel, New Jersey
  - Surgical Studios, Mullica Hill, New Jersey
  - Neptune Surgical Institute, Neptune City, New Jersey
  - Ambulatory Surgical Pavilion at Robert Wood Johnson, New Brunswick, New Jersey
  - RWJ University Hospital - N Brunswick, New Brunswick, New Jersey
  - University Hospital, Newark, New Jersey
  - Specialty Surgical Center of North Brunswick, North Brunswick, New Jersey
  - Global Surgery Center, Oradell, New Jersey
  - North East Regional Surgical Center, Paramus, New Jersey
  - Morris County Surgical Center, Parsippany, New Jersey
  - Capital Health Med Ctr Hopewell, Pennington, New Jersey
  - Chilton Mem Hosp, Pompton Plains, New Jersey
  - Surgical Specialists at Princeton, Princeton, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - MALO Center for Ambulatory Surgery, Rutherford, New Jersey
  - Surgicore of Saddle Brook, Saddle Brook, New Jersey
  - Salem ASC, Salem, New Jersey
  - Hudson Regional Hospital, Secaucus, New Jersey
  - Advanced Surgical Institute, Sewell, New Jersey
  - Jefferson Surgery Center, Sewell, New Jersey
  - Premier Pain Centers, Shrewsbury, New Jersey
  - Shrewsbury Surgery Center, Shrewsbury, New Jersey
  - Jersey Shore Ambulatory Surgery Center, Somers Point, New Jersey
  - Raritan Valley Surgery Center, Somerset, New Jersey
  - Stemmee Surg Ctr, Somerset, New Jersey
  - Univ Ortho Assocs, Somerset, New Jersey
  - University Center for Ambulatory Surgery, Somerset, New Jersey
  - Metropolitan Surgical Institute, South Amboy, New Jersey
  - West Morris Surgery Center, Succasunna, New Jersey
  - Overlook Medical Center, Summit, New Jersey
  - Holy Name Medical Center, Teaneck, New Jersey
  - North Jersey Ortho Spclsts, Teaneck, New Jersey
  - Teaneck Surgery Center, Teaneck, New Jersey
  - The Ctr For Outpatient Surg, Tinton Falls, New Jersey
  - Toms River Surgery Center, Toms River, New Jersey
  - Physicians' SurgiCenter, Toms River, New Jersey
  - Jefferson Washington Twp Hosp, Turnersville, New Jersey
  - Union County Surgery Center, Union, New Jersey
  - Watts Plastic Surgical Center, Vineland, New Jersey
  - St. Joseph's Wayne Hospital, Wayne, New Jersey
  - Advanced Spine and Outpatient Surgery Center, West Orange, New Jersey
  - Mountain Surgery Center, West Orange, New Jersey
  - Pleasantdale Ambulatory Care, West Orange, New Jersey
  - Pascack Valley Medical Center, Westwood, New Jersey
  - Manchester Surgery Center, Whiting, New Jersey
  - Inspira Medical Center, Woodbury, New Jersey
  - TeamMD Surgery Center, Woodland Park, New Jersey
  - Outpatient Surg and Imaging Svcs, Albuquerque, New Mexico
  - University of New Mexico Hospital, Albuquerque, New Mexico
  - VA Medical Center, Albuquerque, New Mexico
  - Modern Pain & Spine PC, Albuquerque, New Mexico
  - Artesia General Hospital, Artesia, New Mexico
  - Everett Road Surgery Center, Albany, New York
  - Amherst Surgery Center, Amherst, New York
  - Auburn Community Hospital, Auburn, New York
  - United Memorial Medical Center, Batavia, New York
  - South Shore Surgery, Bay Shore, New York
  - Southside Hospital, Bay Shore, New York
  - Surgicore North Queens Surgical Center, Bayside, New York
  - Surgicore North Queens, Bayside, New York
  - St. Joseph Hospital, Bethpage, New York
  - Nyu Langone Amb Care Clinic, Brooklyn, New York
  - Brooklyn Surgery Center, Brooklyn, New York
  - Brooklyn VA Medical Center, Brooklyn, New York
  - GoldStep Ambulatory Surgery Center, LLC, Brooklyn, New York
  - NYP -Methodist Hospital, Brooklyn, New York
  - Island Amb Surg Ctr, Brooklyn, New York
  - All City Family Healthcare Center, Brooklyn, New York
  - Allcity Family Hlthcr Ctr, Brooklyn, New York
  - Maimonides Midwood Community Hospital, Brooklyn, New York
  - South Brooklyn Health, Brooklyn, New York
  - ECMC Hospital, Buffalo, New York
  - Atlas Surg Ctr, Buffalo, New York
  - West Surgical ASC, Camillus, New York
  - F.F. Thompson Hospital, Canandaigua, New York
  - Ortho Ny Amb Surg Ctr, Clifton Park, New York
  - Clifton Springs Hospital & Clinic, Clifton Springs, New York
  - OMNI Pain & Precision Medicine, Clinton, New York
  - Noyes Memorial Hospital, Dansville, New York
  - PrecisionCare Surgery Center, East Setauket, New York
  - Specialists One Day Surgery, East Syracuse, New York
  - Ellenville Regional Hospital, Ellenville, New York
  - Arnot Ogden Hospital, Elmira, New York
  - Fishkill Ambulatory Surgery Center, Fishkill, New York
  - Gramercy Surgery Center, Flushing, New York
  - Ainsworth Surgery Center, Garden City, New York
  - NYU Langone ASC - Garden City, Garden City, New York
  - Eastern Long Island Hospital, Greenport, New York
  - Stony Brook Eastern Long Island, Greenport, New York
  - Northway Surgery & Pain Center, Halfmoon, New York
  - Catskill Regional Medical Center, Harris, New York
  - Surgical Specialty Center of Westchester, Harrison, New York
  - Hauppauge SC, Hauppauge, New York
  - Huntington Hospital, Huntington, New York
  - Orthopedic Spine Care of Long Island, Huntington Station, New York
  - Cayuga Medical Center at Ithaca, Ithaca, New York
  - Specialty Surgery Center of CNY, Liverpool, New York
  - Lynbrook Surg Ctr, Lynbrook, New York
  - Crystal Run Healthcare ASC, Middletown, New York
  - Day Op Center of Long Island, Mineola, New York
  - NYU Langone Hospital-Long Island (Winthrop), Mineola, New York
  - ProHealth Ambulatory Surgery Center, New Hyde Park, New York
  - NYU Langone Orthopedic, New York, New York
  - Hudson Medical Group, New York, New York
  - Hudson Surg Ctr, New York, New York
  - VA New York Harbor (Margaret Cochran Corbin Campus), New York, New York
  - Greenwich Village Ambulatory Surgery Center, New York, New York
  - Lenox Health Greenwich Village, New York, New York
  - NYU Ambulatory Care Center, New York, New York
  - NYU Langone Ambulatory Care Center, New York, New York
  - Midtown Surgery Center, New York, New York
  - Surgicare of Manhattan, LLC, New York, New York
  - Surgicore Midtown/Manhattan, New York, New York
  - Manhattan Surgery Center, New York, New York
  - Peak Point Midtown West Asc, New York, New York
  - SurgiCare of Westside, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Fifth Avenue Surgery Center, New York, New York
  - New York Presbyterian Allen Hospital, New York, New York
  - Pain Physician New York, New York, New York
  - Pain Physicians NY, New York, New York
  - Memorial Sloan Kettering, New York, New York
  - Memorial Sloan-Kettering Cancer Center Inc, New York, New York
  - Delmarva Pain, Newark, New York
  - Heritage One Day Surgery, North Syracuse, New York
  - Montefiore Nyack Hospital, Nyack, New York
  - Olean Gen Hosp, Olean, New York
  - Long Island Community Hospital, Patchogue, New York
  - Surgical Pain Center of the Adirondacks, Plattsburgh, New York
  - John T Mather Memorial Hospital, Port Jefferson, New York
  - St Charles Hospital, Port Jefferson, New York
  - Port Jefferson Surgery Center, Port Jefferson Station, New York
  - Nuvance Health Vassar Brothers Medical Center, Poughkeepsie, New York
  - The Surgery Center at Orthopedic Associates LL, Poughkeepsie, New York
  - The Pain Treatment Center - URMC, Rochester, New York
  - Linden Oaks Surgery Center, Rochester, New York
  - Strong Memorial Hospital - University of Rochester, Rochester, New York
  - Mercy Medical Center, Rockville Centre, New York
  - St. Francis Hospital, Roslyn, New York
  - Adirondack Health, Saranac Lake, New York
  - Suffolk Surgery Center, Shirley, New York
  - Phelps Memorial Hospital Center, Sleepy Hollow, New York
  - North Shore Surgi-Center, Smithtown, New York
  - St. Catherine of Siena, Smithtown, New York
  - Richmond Pain Management ASC, Staten Island, New York
  - Richmond University Medical Center, Staten Island, New York
  - Stony Brook Medicine, Stony Brook, New York
  - Stony Brook University Hospital, Stony Brook, New York
  - Specialists One Day Surgery, Syracuse, New York
  - Upstate Univ Hosp, Syracuse, New York
  - Avicenna Surgery Center, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Empire State Ambulatory Surgical Center, The Bronx, New York
  - Omni Surgery Center, Utica, New York
  - Atlantic Surgery Center, West Islip, New York
  - Good Samaritan Hospital, West Islip, New York
  - Apex Surgical Center, Westmoreland, New York
  - Day Op Ctr of Long Island, Woodbury, New York
  - St Johns Riverside Hospital, Yonkers, New York
  - Vidant Roanoke Chowan Hospital- Pain Management, Ahoskie, North Carolina
  - Mission Hospital, Asheville, North Carolina
  - Outpatient Surgery Center of Asheville, Asheville, North Carolina
  - Caromount Partners Llc Dba, Belmont, North Carolina
  - NH Brunswick Medical Center, Bolivia, North Carolina
  - Wakemed Cary Surg Ctr, Cary, North Carolina
  - The Imaging and Spine Center - UNC Hospitals, Chapel Hill, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Novant Health Midtown Outpatient Surgery Center, Charlotte, North Carolina
  - Atrium Health Pineville, Charlotte, North Carolina
  - Charlotte Surgery Center, Charlotte, North Carolina
  - UNC Hospitals - Shared Services, Durham, North Carolina
  - North Carolina Specialty Hospital, Durham, North Carolina
  - CaroMont Regional Medical Center, Gastonia, North Carolina
  - Greensboro Specialty Surgical Center, Greensboro, North Carolina
  - Vidant Medical Center, Greenville, North Carolina
  - Vidant Roanoke-Chowan Hospital Greenville, Greenville, North Carolina
  - Margaret R. Pardee Memorial Hospital, Hendersonville, North Carolina
  - Viewmont Surgery Center, Hickory, North Carolina
  - Premier Surgery Center/Atrium Health Wake Forest Baptist, High Point, North Carolina
  - UNC Hospitals - Hillsborough Campus, Hillsborough, North Carolina
  - Onslow Memorial Hospital, Jacksonville, North Carolina
  - Novant Kernersville Medical Hospital, Kernersville, North Carolina
  - UNC Lenoir Health Care, Kinston, North Carolina
  - Brunswick Surgery Center, Leland, North Carolina
  - Southeastern Ambulatory Surgery Center, LLC, Lumberton, North Carolina
  - Novant Health Matthews Med Ctr, Matthews, North Carolina
  - Carteret General Hospital, Morehead City, North Carolina
  - CarolinaEast Medical Center, New Bern, North Carolina
  - Granville Medical Center, Oxford, North Carolina
  - Firsthealth Moore Regional Hospital, Pinehurst, North Carolina
  - Surgery Center of Pinehurst, Pinehurst, North Carolina
  - Blue Ridge Surgery Center, Raleigh, North Carolina
  - Rex Healthcare, Raleigh, North Carolina
  - Raleigh Neurosurgical and Spine Surgery Center, Raleigh, North Carolina
  - Wake Spine and Specialty Surg Ctr, Raleigh, North Carolina
  - Capital City Surgery Center, Raleigh, North Carolina
  - WakeMed Raleigh Campus, Raleigh, North Carolina
  - Wakemed North Family Health and, Raleigh, North Carolina
  - WakeMed North Hospital, Raleigh, North Carolina
  - Halifax Regional Medical Center, Inc., Roanoke Rapids, North Carolina
  - DLP Rutherford Regional Health System, Rutherfordton, North Carolina
  - EmergeOrtho-Smithfield, Smithfield, North Carolina
  - Johnston Health, Smithfield, North Carolina
  - ECU Health Beaufort Hospital, Washington, North Carolina
  - Wilmington Health ASC, Wilmington, North Carolina
  - Wilmington SurgCare, Wilmington, North Carolina
  - Kimel Park Surgery Center, Winston-Salem, North Carolina
  - NH Medical Park Hospital, Winston-Salem, North Carolina
  - St. Alexius Medical Center, Bismarck, North Dakota
  - Sanford Medical Center, Fargo, North Dakota
  - Center for Pain Medicine and Surgery Center, Fargo, North Dakota
  - North Dakota Surgery Center, Grand Forks, North Dakota
  - Aultman Alliance Community Hospital, Alliance, Ohio
  - UH Samaritan Medical Center, Ashland, Ohio
  - Ashtabula County Medical Center, Ashtabula, Ohio
  - O'Bleness Hospital, Athens, Ohio
  - Cleveland Clinic - Avon Hospital, Avon, Ohio
  - Beachwood Medical Center, Beachwood, Ohio
  - Northern Ohio Surgery Center, Beachwood, Ohio
  - University Hospitals Ahuja Medical Center, Beachwood, Ohio
  - Indu and Raj Soin Medical Center, Beavercreek, Ohio
  - Belpre Distribution Ctr, Belpre, Ohio
  - Brecksville Surgery, Brecksville, Ohio
  - Bucyrus Hospital, Bucyrus, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Dcr Surgery Center, Llc, Centerville, Ohio
  - DCR Surgery Center, Centerville, Ohio
  - Miami Valley South Hospital, Centerville, Ohio
  - Adena Health System, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - VA Medical Center Cincinnati, Cincinnati, Ohio
  - Jewish Hospital - Mercy Health, Cincinnati, Ohio
  - JourneyLite of Cincinnati, Cincinnati, Ohio
  - TriHealth Evendale Hospital, Cincinnati, Ohio
  - Bethesda Orthopedic Surgery Center, Cincinnati, Ohio
  - Mercy Anderson Asc, Cincinnati, Ohio
  - Mercy Hosp Anderson Hosp, Cincinnati, Ohio
  - Bethesda North Hospital, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - VA Medical Center Cleveland, Cleveland, Ohio
  - Metro Main Campus, Cleveland, Ohio
  - Metro Health and Surgery Center, Cleveland, Ohio
  - Metrohealth West 150th Health and, Cleveland, Ohio
  - Cleveland Clinic - Pain Management, Cleveland, Ohio
  - SRMC Surg and Outpatient Pavilion, Columbiana, Ohio
  - Ohio State East Hospital, Columbus, Ohio
  - Taylor Station Surgical Center, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Gemini Surgery Center, Columbus, Ohio
  - Lake Health TriPoint Medical Center, Concord, Ohio
  - Univ Hosps Conneaut Medic, Conneaut, Ohio
  - Western Reserve Hospital, Cuyahoga Falls, Ohio
  - Riverview Health Institute, Dayton, Ohio
  - Miami Valley Ambulatory Surgery Center, Dayton, Ohio
  - Surgery Center at Corporate Way, Dayton, Ohio
  - Bradenton Surgery Center, Dublin, Ohio
  - Dublin Surgery Center, Dublin, Ohio
  - Miami Valley Hospital North, Englewood, Ohio
  - Fairfield Hospital, Fairfield, Ohio
  - Galion Community Hospital, Galion, Ohio
  - Holzer Gallipolis, Gallipolis, Ohio
  - Univ Hosps Geneva Med Ctr, Geneva, Ohio
  - Adena Greenfield Medical Center, Greenfield, Ohio
  - Fort Hamilton Hospital, Hamilton, Ohio
  - Highland District Hospital, Hillsboro, Ohio
  - Lancaster Specialty Surgery Center, Lancaster, Ohio
  - Precision Pain care, Lancaster, Ohio
  - Hocking Valley Community Hospital, Logan, Ohio
  - Lorain Surgery Center, Lorain, Ohio
  - Mercy Regional Medical Center, Lorain, Ohio
  - Selby Gen Hosp, Marietta, Ohio
  - Marion Med Cmps, Marion, Ohio
  - New Horizons Surgery Center, Marion, Ohio
  - Southwest Ohio Pain Management Ambulatory Surgery Center, Mason, Ohio
  - Hillcrest Hospital, Mayfield Heights, Ohio
  - Lake County Pain & Diagnostic Center LLC, Mentor, Ohio
  - Mentor Surgery Center, Mentor, Ohio
  - Sycamore Hospital, Miamisburg, Ohio
  - Atrium Medical Center, Middletown, Ohio
  - Southwest Ohio Surgery Center, Middletown, Ohio
  - Fisher-Titus Medical Center, Norwalk, Ohio
  - Mercy Health Allen Hosp, Oberlin, Ohio
  - Mercy St. Charles Hospital, Oregon, Ohio
  - West Central Surgical Center Bayside, Oregon, Ohio
  - Aultman Orville, Orrville, Ohio
  - MetroHealth Parma Medical Center, Parma, Ohio
  - Three Gables Surgery Center, Proctorville, Ohio
  - UH Portage Medical Center, Ravenna, Ohio
  - Salem Cmnty Hosp, Salem, Ohio
  - Erie Shores Surg Ctr, Sandusky, Ohio
  - University Hospitals- Suburban, South Euclid, Ohio
  - Ohio Valley Surgical Hospital, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - The University of Toledo Medical Center, Toledo, Ohio
  - Deca Health, Toledo, Ohio
  - West Central Surgical Center, Toledo, Ohio
  - St. Anne Hospital, Toledo, Ohio
  - Toledo Clinic Outpatient Surgery, Toledo, Ohio
  - Cleveland Clinic - Twinsburg Family Health & Surgery Center, Twinsburg, Ohio
  - St. Mina Interventional Pain Center, Warren, Ohio
  - Trumbull Regional Medical Center, Warren, Ohio
  - St Joseph Pain Mgmt Ctr, Warren, Ohio
  - Adena Pike Medical Center, Waverly, Ohio
  - West Chester Surgical Suites, West Chester, Ohio
  - Eastwind Surgical LLC, Westerville, Ohio
  - University Hospitals Health System St John Medical Center, Westlake, Ohio
  - Lake Health West Med Ctr, Willoughby, Ohio
  - Great Lakes Pain Management, Willoughby Hills, Ohio
  - Wright Patterson Hospital, Wright-Patterson Air Force Base, Ohio
  - The Orthopedic Surgery Center, Youngstown, Ohio
  - Youngstown Orthopedic Associates, Youngstown, Ohio
  - Genesis Hosp, Zanesville, Ohio
  - Apex Surgery Center, Ada, Oklahoma
  - Ardmore Regional Surgery Center, Ardmore, Oklahoma
  - Mercy Hospital Ardmore, Ardmore, Oklahoma
  - Grady Memorial Hosp, Chickasha, Oklahoma
  - Southern Plains Med Ctr, Chickasha, Oklahoma
  - Duncan Regional Hospital, Duncan, Oklahoma
  - Summit Medical Center, Edmond, Oklahoma
  - Pain & Sleep Institute of Oklahoma, Edmond, Oklahoma
  - Great Plains Regional Medical Center, Elk City, Oklahoma
  - St Marys Regional Med Ctr, Enid, Oklahoma
  - Surgery Center of Enid, Enid, Oklahoma
  - Eastern Oklahoma Va Health Care, Muskogee, Oklahoma
  - St Anthony Hospital, Oklahoma City, Oklahoma
  - OneCore Health, Oklahoma City, Oklahoma
  - Oklahoma Spine Surgery Center, Oklahoma City, Oklahoma
  - Oklahoma Pain Physicians, Oklahoma City, Oklahoma
  - Surgical Hospital of Oklahoma, Oklahoma City, Oklahoma
  - Mem Pain Surg Ctr, Oklahoma City, Oklahoma
  - Oklahoma Heart Hosp South, Oklahoma City, Oklahoma
  - OCOM South, Oklahoma City, Oklahoma
  - OCOM North, Oklahoma City, Oklahoma
  - Tulsa Amb Procedure, Tulsa, Oklahoma
  - Oklahoma State University Medical Center, Tulsa, Oklahoma
  - Tulsa Procedure Suites, Tulsa, Oklahoma
  - Waverly Surgery Center, Albany, Oregon
  - Saint Alphonsus Medical Center Baker City, Baker City, Oregon
  - Cornell Surgery Center, Beaverton, Oregon
  - Oregon Surgical Institute, Beaverton, Oregon
  - Bend Surgery Center, Bend, Oregon
  - Central Oregon Surgical Institute, Bend, Oregon
  - Deschutes Surgery Center, Bend, Oregon
  - Chase Gardens Surgery Center, Eugene, Oregon
  - Two Rivers Surgical Center, Eugene, Oregon
  - Burnside Surgery Center, Gresham, Oregon
  - Good Shepherd Medical Center, Hermiston, Oregon
  - Crater Lake Surgery Center, Medford, Oregon
  - Columbia Pain Management, PC, Milwaukie, Oregon
  - Saint Alphonsus Medical Center Ontario, Ontario, Oregon
  - East Portland Surgery Center, Portland, Oregon
  - Pearl Womens Ctr, Portland, Oregon
  - Oregon Pain Center, Portland, Oregon
  - Oregon Specialists Surgery Center, Salem, Oregon
  - Pacific Northwest Surgery Center, Springfield, Oregon
  - Oregon Outpatient Surgery Center, Tigard, Oregon
  - Cascade Spine Center, Tualatin, Oregon
  - South Portland Surgical Center, Tualatin, Oregon
  - Northwest Spine and Laser Surgery Center, Wilsonville, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Carepath Injury Ctr of Pennsylvania, Allentown, Pennsylvania
  - Cedar Crest Surg Ctr, Allentown, Pennsylvania
  - Lehigh Valley Hospital - Cedar Crest, Allentown, Pennsylvania
  - Surgery Center of Allentown, Allentown, Pennsylvania
  - Allegheny Surgery Center, Altoona, Pennsylvania
  - Ctr For the Surgl Arts, Altoona, Pennsylvania
  - Ambulatory Surgery Center of Bala Cynwyd, Bala-Cynwyd, Pennsylvania
  - Bethel Park Surgery Center, Bethel Park, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Center for Specialized Surgery LP, Bethlehem, Pennsylvania
  - Valley Surgical Ctr, Bethlehem, Pennsylvania
  - Susquehanna Surgery Center, Bloomsburg, Pennsylvania
  - Radiance Surgery Center, Bridgeville, Pennsylvania
  - Bryn Mawr Orthopedic Surgery Center, Bryn Mawr, Pennsylvania
  - Bucks County Surgl Suites Highpoint, Chalfont, Pennsylvania
  - New Britain Surgery Center, Chalfont, Pennsylvania
  - St. Luke's Miners Campus, Coaldale, Pennsylvania
  - Brandywine Hospital, Coatesville, Pennsylvania
  - Lehigh Valley Hosp Dickson City, Dickson City, Pennsylvania
  - Einstein Medical Center Montgomery, East Norriton, Pennsylvania
  - Lehigh Valley Hospital - Hecktown, Easton, Pennsylvania
  - Greater Erie Surgery Center, LLC, Erie, Pennsylvania
  - Greater Erie Surgery Center, Erie, Pennsylvania
  - The Surgery Center of Chester County, Exton, Pennsylvania
  - The Surgery Center at Fort Washington, Fort Washington, Pennsylvania
  - AHN Grove City, Grove City, Pennsylvania
  - Grand View Surgery Center at Harleysville, Harleysville, Pennsylvania
  - Susquehanna Valley Pain Management, Harrisburg, Pennsylvania
  - Hershey Outpatient Surgery Center, Hershey, Pennsylvania
  - Milton S Hershey Medical Center, Hershey, Pennsylvania
  - FSA of Huntingdon Valley, LLC, Huntingdon Valley, Pennsylvania
  - Valley Pain Center, Huntingdon Valley, Pennsylvania
  - Indiana Regional Medical Center, Indiana, Pennsylvania
  - Main Line Spine Surgery Center, King of Prussia, Pennsylvania
  - Riverview Ambulatory Surgical Center, Kingston, Pennsylvania
  - Lancaster Gen Health, Lancaster, Pennsylvania
  - Surgery Center of Lancaster, L.P., Lancaster, Pennsylvania
  - Advanced Surgery Center of Lancaster, Lancaster, Pennsylvania
  - Forest Health Medical Center of Bucks County, Langhorne, Pennsylvania
  - Langhorne Surgical Center, Langhorne, Pennsylvania
  - Lansdale Hospital, Lansdale, Pennsylvania
  - Montgomery Surgery Center, Lansdale, Pennsylvania
  - North Pointe Surg Ctr, Lebanon, Pennsylvania
  - Physicians Surgical Center, Lebanon, Pennsylvania
  - Integrated Surgical Institute, Leesport, Pennsylvania
  - Lehigh Valley Hospital-Carbon, Lehighton, Pennsylvania
  - Ohio Valley Hospital, McKees Rocks, Pennsylvania
  - Meadville Medical Center, Meadville, Pennsylvania
  - Penn Highlands Mon Valley, Monongahela, Pennsylvania
  - Spartan Health Surgicenter, Monongahela, Pennsylvania
  - Forbes Hosp, Monroeville, Pennsylvania
  - Geisinger Med Ctr Muncy, Muncy, Pennsylvania
  - Philadelphia Surgical Center, Narberth, Pennsylvania
  - Penn Presbyterian Med Ctr, Philadelphia, Pennsylvania
  - Presbyterian Medical Center, Philadelphia, Pennsylvania
  - Philadelphia Pain, Philadelphia, Pennsylvania
  - Thomas Jefferson Univ Hosp, Philadelphia, Pennsylvania
  - Jefferson Surgical Center at the Navy Yard, Philadelphia, Pennsylvania
  - Gabay and Gottlief Cosmetic Surg Ct, Philadelphia, Pennsylvania
  - Philadelphia Surgi Center, Philadelphia, Pennsylvania
  - Chestnut Hill Hospital, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Penn Med At Rittenhouse, Philadelphia, Pennsylvania
  - Jefferson Methodist Hospital, Philadelphia, Pennsylvania
  - West Penn Hosp, Pittsburgh, Pennsylvania
  - Gamma Surgery Center, Pittsburgh, Pennsylvania
  - Northeast Regional Surgery Center, Plains, Pennsylvania
  - PMSI - Pain Medicine Divison, Pottstown, Pennsylvania
  - Pottstown Hospital, Pottstown, Pennsylvania
  - Lehigh Valley Hospital-Schuylkill, Pottsville, Pennsylvania
  - Premier Pain Professionals (Tilden Surgery Center), Pottsville, Pennsylvania
  - Penn Medicine Radnor, Radnor, Pennsylvania
  - North East Surgery Center, Scranton, Pennsylvania
  - Somerset Community Hospital, Somerset, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - St Lukes Hosp Monroe CMPS, Stroudsburg, Pennsylvania
  - Edgewood Surgical Hospital, Transfer, Pennsylvania
  - Trevose Specialty Care Surgical Center, Trevose, Pennsylvania
  - Warren General Hospital, Warren, Pennsylvania
  - Bucks County Surgical Suites, Warrington, Pennsylvania
  - South Hills Surgery Center, West Mifflin, Pennsylvania
  - Western PA Surgery Center, Wexford, Pennsylvania
  - Interventional & Surgical Suites of Wilkes - Barre, LLC, Wilkes-Barre, Pennsylvania
  - Wilkes Barre General Hospital, Wilkes-Barre, Pennsylvania
  - Pain Center of Wyoming Valley, LLC, Wilkes-Barre Township, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Surgical Institute of Reading, Wyomissing, Pennsylvania
  - Wyomissing Surgical Services, Wyomissing, Pennsylvania
  - OSS Health Powder Mill, York, Pennsylvania
  - Crossings Surgery Center, Warwick, Rhode Island
  - Aiken Regional Medical Center, Aiken, South Carolina
  - Med Univ Hosp Autg, Charleston, South Carolina
  - MUSC Rutledge Tower, Charleston, South Carolina
  - Palmetto Health USC Medical Group, Columbia, South Carolina
  - MUSC Health Columbia Medical Center Downtown, Columbia, South Carolina
  - William Jennings Bryan Dorn Va Med, Columbia, South Carolina
  - Atlantic Coast Pain Specialists, Conway, South Carolina
  - Rivertown Surgery Center, Conway, South Carolina
  - The Surgery Center at Edgewater, Fort Mill, South Carolina
  - Piedmont Surgery Center, Greenville, South Carolina
  - Summit Spine and Joint Ctr, Greenville, South Carolina
  - Coastal Carolina Hospital, Hardeeville, South Carolina
  - Center for Advanced Surgery, Ladson, South Carolina
  - McLeod Seacoast OR, Little River, South Carolina
  - East Cooper Medical Center, Mt. Pleasant, South Carolina
  - Signe Spine Surgl Ctr, Mt. Pleasant, South Carolina
  - Southeastern Spine Institute ASC, Mt. Pleasant, South Carolina
  - Southern Grace Pain and Regenerative Medicine, Mt. Pleasant, South Carolina
  - Parkway Surgery Center, Myrtle Beach, South Carolina
  - Bluffton Okatie Outpatient Center, Okatie, South Carolina
  - Prisma Health-Upstate - Materials Distribution Center, Simpsonville, South Carolina
  - Ambulatory Surgery Center of Spartanburg, Spartanburg, South Carolina
  - Palmetto Health Toumey, Sumter, South Carolina
  - Brookings Ambulatory Surgery Center, Brookings, South Dakota
  - Milbank Area Hosp Avera Health, Milbank, South Dakota
  - Plastic Surgical Center of Rapid City, Rapid City, South Dakota
  - Same Day Surgery Center, Rapid City, South Dakota
  - Black Hills Surgical Hospital, Rapid City, South Dakota
  - Monument Health Rapid City Hospital, Rapid City, South Dakota
  - Innovative Procedural Center, Watertown, South Dakota
  - Saint Francis Hospital-Bartlett, Bartlett, Tennessee
  - Crossroads Surgery Center, Brentwood, Tennessee
  - Bristol Regional Medical Center, Bristol, Tennessee
  - Riverfront Surgery Center, Chattanooga, Tennessee
  - Center for Sports Medicine and Orthopaedics Ambulatory Surgery Center, Chattanooga, Tennessee
  - Parkridge Medical Center, Chattanooga, Tennessee
  - Ipc Surg Ctr, Cleveland, Tennessee
  - The Surgery Center of Cleveland, Cleveland, Tennessee
  - Surg Ctr of Mid Tennessee, Columbia, Tennessee
  - Cookeville Regional Medical Center (N Washington Ave), Cookeville, Tennessee
  - Spectrum Pain Clinic, Cordova, Tennessee
  - Cool Springs Surgery Center LLC, Franklin, Tennessee
  - Summit Surgery Center, Hermitage, Tennessee
  - Chattanooga Pain Surgery Center, Hixson, Tennessee
  - Midsouth Interventional Pain, Jackson, Tennessee
  - Physicians Surgery Center/Jackson, Jackson, Tennessee
  - Spectrum Pain Clinic, Jackson, Tennessee
  - Physician's Surgery Center of Knoxville, Knoxville, Tennessee
  - Turkey Creek Medical Center (Tennova), Knoxville, Tennessee
  - Blount Mem Hosp, Maryville, Tennessee
  - Prisma Health Outpatient Surgery, Maryville, Tennessee
  - Medical Education and Research Institute, Memphis, Tennessee
  - Mays and Schnapp Neurospine and, Memphis, Tennessee
  - Providence Surgery Center, Mount Juliet, Tennessee
  - James H Quillen Va Med Ctr, Mountain Home, Tennessee
  - Premier Orthopaedic Surgery Center - Nashville, Nashville, Tennessee
  - Methodist Medical Center, Oak Ridge, Tennessee
  - Spine and Pain Physicians Surgery Center, Smyrna, Tennessee
  - Southern Tennessee Reg Health, Winchester, Tennessee
  - Abilene Ctr For Ortho and Multi, Abilene, Texas
  - Abilene Spine and Joint Surgery Center, Abilene, Texas
  - Hendrick Med Ctr South, Abilene, Texas
  - Ambulatory Surgical Institute of Dallas, Addison, Texas
  - Northaven Surg Ctr, Allen, Texas
  - Surgery Center of Amarillo, Amarillo, Texas
  - Acute & Chronic Pain and Spine Center Ambulatory Surgery Center, Amarillo, Texas
  - Memorial Hermann Surgery Center Brazoria, Angleton, Texas
  - Legent Outpatient Surgery Austin, Austin, Texas
  - Orthopaedic Associates of Central Texas Surgery Center, LLC, Austin, Texas
  - Falconhead Surgery Center, Austin, Texas
  - South Austin Surgery Center, Austin, Texas
  - Stonegate Surgery Center, Austin, Texas
  - PSA Ambulatory Surgical Center of South Austin, LLC, Austin, Texas
  - Water Leaf Surgery Center, LTD, Austin, Texas
  - Spicewood Surg Ctr, Austin, Texas
  - Capitol Pain Institute, Austin, Texas
  - Center for Specialty Surgery of Austin, Austin, Texas
  - PSA Ambulatory Surgical Center of Austin, LLC, Austin, Texas
  - Altus Baytown Hospital, Baytown, Texas
  - Baytown Hospital, Baytown, Texas
  - Baytown Medical Center, Baytown, Texas
  - Houston Methodist Baytown Hospital, Baytown, Texas
  - Houston Methodist Surgery Center, Baytown, Texas
  - CHRISTUS Southeast Texas -St. Elizabeth, Beaumont, Texas
  - Riceland Surgery Center, Beaumont, Texas
  - The Medical Center of Southeast Texas-Beaumont Campus, Beaumont, Texas
  - Advanced Surgical Care of Boerne, Boerne, Texas
  - St. Joseph Health Regional Hospital - Bryan, Bryan, Texas
  - Legent Orthopedic Hospital, Carrollton, Texas
  - Carrollton Reg Med Ctr, Carrollton, Texas
  - Castle Hills Surgicare, Carrollton, Texas
  - Amc Cavazos - Pa, Cavazos, Texas
  - Cedar Park Surgery Center, Cedar Park, Texas
  - Baylor Scott & White College Station Hospital, College Station, Texas
  - St Joseph College Station, College Station, Texas
  - Columbus Community Hosp, Columbus, Texas
  - North Pines Surgery Center, Conroe, Texas
  - VIP Surgical Center, Conroe, Texas
  - Legent Institute of Specialized Surgery, Conroe, Texas
  - Saratoga Surgical Center, Corpus Christi, Texas
  - Spinecare, Corpus Christi, Texas
  - Texas Precision Surgery Center, Corpus Christi, Texas
  - Texas Ortho Ctr of Excellence, Corpus Christi, Texas
  - Houston Meth Cypress Hosp, Cypress, Texas
  - Horizon Medical Center, Dallas, Texas
  - Dallas Medical Center, Dallas, Texas
  - Univ of Texas Southwestern Med Ctr, Dallas, Texas
  - Utsw Zale Lipshy, Dallas, Texas
  - Montfort Surgery Center, Dallas, Texas
  - Baylor Scott and White Surgicare, Dallas, Texas
  - Baylor Scott & White Surgicare North Dallas, Dallas, Texas
  - Premier Pain Solutions, Dallas, Texas
  - WHS East Campus, Decatur, Texas
  - STHS - Edinburg Hospital, Edinburg, Texas
  - Advanced Surg Ctr of El Paso, El Paso, Texas
  - El Paso Center for GI, El Paso, Texas
  - El Paso Specialty Hospital, El Paso, Texas
  - Sierra Medical Center, El Paso, Texas
  - Gateway Surgical Center, El Paso, Texas
  - Physicians West El Paso Surg Ctr, El Paso, Texas
  - Advancedcare Surg Ctr, Ennis, Texas
  - Carl R Darnall Army Med Ctr, Fort Cavazos, Texas
  - Baylor Surgicare at Fort Worth, Fort Worth, Texas
  - John Peter Smith Hosp, Fort Worth, Texas
  - Baylor Scott & White Surgical Hospital at Fort Worth, Fort Worth, Texas
  - Preston Surg Ctr, Frisco, Texas
  - Coryell Health, Gatesville, Texas
  - Glen Rose Med Ctr, Glen Rose, Texas
  - Granbury Hosp Corp, Granbury, Texas
  - Hamilton Gen Hosp, Hamilton, Texas
  - Optimum Pain & Regenerative Medicine, Harlingen, Texas
  - Platinum Surgery Center, Harlingen, Texas
  - SportsOrtho Surg Ctr, Harlingen, Texas
  - Museum District Ambulatory Surgery Center, Houston, Texas
  - Memorial Hermann Surgery Center Greater Heights, Houston, Texas
  - The Heights Hospital, Houston, Texas
  - Complete Surgery Center Northwest, Houston, Texas
  - Houston Premier Surgery Center in The Villages, Houston, Texas
  - Memorial Ambulatory Surgery Center, Houston, Texas
  - Memorial Hermann West Houston Surgery Center, Houston, Texas
  - Townsen Memorial ASC Medical Center, Houston, Texas
  - River Oaks Hospital and Clinics, Houston, Texas
  - Baylor College of Medicine Med Ctr, Houston, Texas
  - Memorial Hermann Surgery Center - Main Street, Houston, Texas
  - Memorial Hermann Surgery Center Main Street, Houston, Texas
  - U.T MD Anderson Cancer Center, Houston, Texas
  - Inov8 Orthopedics, Houston, Texas
  - Memorial Hermann Surgery Center Memorial Village, Houston, Texas
  - University Pain Associates, Houston, Texas
  - East Houston Medical Center, Houston, Texas
  - Houston Surgery Center, Houston, Texas
  - Innovative Solutions, LLC, Houston, Texas
  - Memorial Houston Surgery Center, Houston, Texas
  - Body Balance Chiropractic and Wellness, Houston, Texas
  - Houston Methodist Orthopedic & Sports Medicine, Houston, Texas
  - Houston Methodist Willowbrook Hospital, Houston, Texas
  - Altus Houston Hospital, Houston, Texas
  - Crystal Outpatient Surgery Center, Houston, Texas
  - Hca Houston Hlthcr Northwest, Houston, Texas
  - Memorial Hermann Surgery Center North Houston Endoscopy and Surgery, Houston, Texas
  - Northwest Surg Ctr Red Oak, Houston, Texas
  - TOPS Specialty Hospital, Houston, Texas
  - United Memorial Medical Center - North Hospital, Houston, Texas
  - Paramount Surgical Center, Houston, Texas
  - Spring Hospital, Houston, Texas
  - Brooke Army Medical Center, Houston, Texas
  - Humble Vascular Surgical Center, Humble, Texas
  - Townsen Memorial Hospital, Humble, Texas
  - Townsen Mem Surg Ctr Katy, Katy, Texas
  - Houston Orthopedic and Spine Surgery Center, Katy, Texas
  - Memorial Hermann Surgery Center - Kingsland, Katy, Texas
  - Bear Creek Surg Ctr, Keller, Texas
  - Ambulatory Surgery Center of Killeen, Killeen, Texas
  - Central Texas Day Surgery Center, Killeen, Texas
  - AdventHealth Central Texas, Killeen, Texas
  - Memorial Hermann Specialty Hosp, Kingwood, Texas
  - Townsen Memorial Surgery Center-Kingwood, Kingwood, Texas
  - Hays Surgery Center, Kyle, Texas
  - Plum Creek Surgery Center LLC, Kyle, Texas
  - Laredo Medical Center, Laredo, Texas
  - Doctors Hospital of Laredo, Laredo, Texas
  - UTMB Health League City Campus Hospital, League City, Texas
  - Advanced Pain Institute of Texas, Lewisville, Texas
  - Seva Pain and Wellness, Lewisville, Texas
  - CHRISTUS Good Shepherd Medical Center - Longview, Longview, Texas
  - Longview Reg Med Ctr, Longview, Texas
  - Grace Medical Center - OP, Lubbock, Texas
  - Lubbock Surg Ctr, Lubbock, Texas
  - Grace Medical Center, Lubbock, Texas
  - Woodland Heights Med Center, Lufkin, Texas
  - Baylor Scott & White Medical Center - Marble Falls, Marble Falls, Texas
  - Valley Ambulatory Surgery Center, McAllen, Texas
  - Glatz Group, McAllen, Texas
  - Baylor Scott and White Med Ctr, McKinney, Texas
  - NTTC Surgery Center, Mesquite, Texas
  - Upper Valley Dialysis ASC, Mission, Texas
  - Titus County Mem Hosp, Mount Pleasant, Texas
  - Houston Methodist Clear Lake Hospital, Nassau Bay, Texas
  - Christus Physicians Ambulatory Surgery Center, New Braunfels, Texas
  - New Braunfels Surgery Center, New Braunfels, Texas
  - Altus Pasadena Surgical Center, Pasadena, Texas
  - Chi St Lukes Health Patience Med, Pasadena, Texas
  - Doctors United Surgery Center, Pasadena, Texas
  - Austin Oral Surg, Pflugerville, Texas
  - Baylor Scott & White Surgicare at Plano Alliance, Plano, Texas
  - Star Med Ctr, Plano, Texas
  - Peak Health Surgicare of Horizon Medical Center, Richardson, Texas
  - Texas Health Surg Ctr Rockwall, Rockwall, Texas
  - Babcock Surgical Center, San Antonio, Texas
  - First Choice Asc, San Antonio, Texas
  - St. Luke's Baptist Hospital, San Antonio, Texas
  - Univ Hosp, San Antonio, Texas
  - Ut Health Marc Asc, San Antonio, Texas
  - Univ Health Surg Ctr Mac, San Antonio, Texas
  - San Antonio Military Med Ctr, San Antonio, Texas
  - Foundation Hospital, San Antonio, Texas
  - Legent Orthopedic and Spine, San Antonio, Texas
  - Christus Santa Rosa Hosp Westover, San Antonio, Texas
  - Legent Westover Hills Surgery Center, San Antonio, Texas
  - North Central Baptist Hospital, San Antonio, Texas
  - Advanced Surgery Center of San Antonio, LLC, San Antonio, Texas
  - Memorial Hermann Surg Ctr the Woodlands, Shenandoah, Texas
  - Houston Methodist The Woodlands Hospital, Shenandoah, Texas
  - North Texas Surgery Center, Sherman, Texas
  - Castle Surg Ctr, Southlake, Texas
  - Medical City Surgery Center Southlake, Southlake, Texas
  - WHS Pain Management Center at Southlake, Southlake, Texas
  - Advanced Spine and Pain Specialists, Spring, Texas
  - Preva Surgicare, Spring, Texas
  - Townsen Memorial Surgery Center Spring, Spring, Texas
  - Spring Hospital, Spring, Texas
  - Sugar Land Surg Ctr, Sugar Land, Texas
  - United Memorial Medical Center, Sugar Land, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Memorial Hermann Surgical Hospital First Colony, Sugar Land, Texas
  - One Step Diagnostic Sugar Land, Sugar Land, Texas
  - Christus Mother Frances Hospital, Sulphur Springs, Texas
  - Baylor Scott & White Medical Center Sunnyvale, Sunnyvale, Texas
  - Baylor Scott and White Pain Clinic, Temple, Texas
  - Christus St Michael Health System, Texarkana, Texas
  - Precision Surg Ctr, Texarkana, Texas
  - MHSC Woodlands Parkway, The Woodlands, Texas
  - Alpha Surgery Center, Tomball, Texas
  - Executive Surgery Center, Tomball, Texas
  - Legent North Houston Surgical Hospital, Tomball, Texas
  - Cataract Center of East Texas, Tyler, Texas
  - Texas Spine & Joint Hospital, Tyler, Texas
  - Tyler Tx Asc, Tyler, Texas
  - Trinity Mother Frances Hospital, Tyler, Texas
  - Christus Surgery Center at Olympia Hills, Universal City, Texas
  - Citizens Medical Center, Victoria, Texas
  - DeTar Hospital North, Victoria, Texas
  - The Surgery Center, Victoria, Texas
  - Texas Pain Physicians, Waxahachie, Texas
  - Houston Physicians Hospital, Webster, Texas
  - University of Texas Medical Branch - Clear Lake, Webster, Texas
  - Rio Grande Pain Team, Weslaco, Texas
  - Precision Regenerative and Functional Medicine, West Lake Hills, Texas
  - Maplewood Ambulatory Surgery Center, Wichita Falls, Texas
  - Advanced Surg Ctr of Northern Utah, Logan, Utah
  - Cache Valley Surg Ctr, Logan, Utah
  - Southwest Spine and Pain Ctr, Logan, Utah
  - Moab Regional Hospital, Moab, Utah
  - Vineyard Surg Ctr, Orem, Utah
  - Global Microsurgical Ctr of Park, Park City, Utah
  - Castleview Hospital, Price, Utah
  - Spring Creek Surgical Center, Providence, Utah
  - Uintah Basin Medical Center, Roosevelt, Utah
  - Intermountain Surg Ctr Tosh, Salt Lake City, Utah
  - Surg Ctr At South Ogden, South Ogden, Utah
  - Coral Desert Surgery Center LLC, St. George, Utah
  - Zion Eye Institute, St. George, Utah
  - Northpointe Surgical Ctr, Tooele, Utah
  - Jordan Valley Hosp, West Jordan, Utah
  - Holy Cross Hosp Jordan Valley West, West Valley City, Utah
  - Jordan Valley Med Ctr West Valley, West Valley City, Utah
  - Fletcher Allen Hlthcr, Williston, Vermont
  - Univ of Vermont Med, Williston, Vermont
  - Monticello Community Surgery Center, Charlottesville, Virginia
  - University of Virginia Health System, Charlottesville, Virginia
  - Uva Med Ctr 29 Warehouse, Charlottesville, Virginia
  - New River Valley Surg Ctr, Christiansburg, Virginia
  - Fairfax Surgical Ctr, Fairfax, Virginia
  - Spine and Pain Clinics of North, Fairfax, Virginia
  - Augusta Health, Fishersville, Virginia
  - Sentara RMH Medical Center, Harrisonburg, Virginia
  - Haymarket Surgery Center, Haymarket, Virginia
  - VCU Health Ambulatory Surgery Center, Henrico, Virginia
  - Virginia Commonwealth Univ, Henrico, Virginia
  - Surgery Center of Lynchburg, Lynchburg, Virginia
  - Prince William Surgery Center, Manassas, Virginia
  - The Spine Care, Manassas, Virginia
  - National Spine and Pain Centers, McLean, Virginia
  - Johnston Willis Hospital, North Chesterfield, Virginia
  - Southside Regional Med Ctr, Petersburg, Virginia
  - Capital Spine and Pain Ctrs, Reston, Virginia
  - Virginia Spine Instu, Reston, Virginia
  - Hunter Holmes McGuire VA Med Ctr, Richmond, Virginia
  - Chippenham Hospital, Richmond, Virginia
  - Henrico Doctors Hospital, Richmond, Virginia
  - Johnston Willis Hosp, Richmond, Virginia
  - VA Medical Center Richmond, Richmond, Virginia
  - VCU Health System Authority, Richmond, Virginia
  - Virginia Interventional Pain and, Roanoke, Virginia
  - Blue Ridge Surgery Center, Salem, Virginia
  - Lewis Gale Hospital, Salem, Virginia
  - Valley Health Surgery Center, Winchester, Virginia
  - Island Health Hospital, Anacortes, Washington
  - Anesis Pain- Bel-Red ASC, Bellevue, Washington
  - Bellevue Surgery Center, Bellevue, Washington
  - Mt. Baker Surgery Center, Bellingham, Washington
  - Tri-State Memorial Hospital, Clarkston, Washington
  - Proliance Eastside Surgery Center, Kirkland, Washington
  - Samaritan Healthcare, Moses Lake, Washington
  - Olympia Surg Ctr, Olympia, Washington
  - Pacific Surgery Center, Poulsbo, Washington
  - Prosser Memorial Hospital, Prosser, Washington
  - Proliance Surgery Center, Renton, Washington
  - Apex Spine Institute ASC, Richland, Washington
  - Puget Sound Pain Clinic, Tukwila, Washington
  - The Vancouver Clinic Inc., Vancouver, Washington
  - Raleigh Gen Hosp, Beckley, West Virginia
  - Raleigh General Hospital, Beckley, West Virginia
  - The Saint Francis Hospital Center for Pain Relief, Charleston, West Virginia
  - Day Surgery Center, Charleston, West Virginia
  - Davis Medical Center, Elkins, West Virginia
  - Cabell Huntington Hospital, Huntington, West Virginia
  - St Marys Med Ctr, Huntington, West Virginia
  - Charleston Area Med Ctr Teays, Hurricane, West Virginia
  - Logan Regional Medical Center, Logan, West Virginia
  - Tri-State Surgical Center, Martinsburg, West Virginia
  - WV University Hospitals, Morgantown, West Virginia
  - Wetzel County Hospital, New Martinsville, West Virginia
  - Camden Clark Medical Center, Parkersburg, West Virginia
  - Jackson General Hospital, Ripley, West Virginia
  - Thomas Mem Hosp, South Charleston, West Virginia
  - Roane General Hospital, Spencer, West Virginia
  - Wheeling Hospital, Wheeling, West Virginia
  - Oakleaf Surgl Hosp, Altoona, Wisconsin
  - ThedaCare Medical Center - Orthopedic Spine & Pain, Appleton, Wisconsin
  - ThedaCare Regional Medical Center-Appleton, Appleton, Wisconsin
  - Mayo Clinic Health System Northland, Barron, Wisconsin
  - Aurora Health Center Southern Lakes, Burlington, Wisconsin
  - Aurora St Lukes South Shore, Cudahy, Wisconsin
  - Upland Hills Health, Dodgeville, Wisconsin
  - Oakleaf Surgical Hosp, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Eau Claire, Eau Claire, Wisconsin
  - Edgerton Hospital and Health Services, Edgerton, Wisconsin
  - Aurora Health Care Southern Lakes, Inc.- Elkhorn, Elkhorn, Wisconsin
  - Aurora Health Fond Du Lac, Fond du Lac, Wisconsin
  - Milwaukee Surgical Suites LLC, Franklin, Wisconsin
  - Neurosurgery and Endovascular Associates LLC, Franklin, Wisconsin
  - The Surgery Center LLC, Franklin, Wisconsin
  - Geneva Surgical Suites LLC, Genoa City, Wisconsin
  - AHCMG Sugery Center Germantown, Germantown, Wisconsin
  - Aurora Germantown, Germantown, Wisconsin
  - Bellin Memorial Hospital, Green Bay, Wisconsin
  - Aurora Baycare Medical Center-Discovery, Green Bay, Wisconsin
  - Aurora Baycare Medical Center, Green Bay, Wisconsin
  - Spine Solutions of Green Bay, LLC, Green Bay, Wisconsin
  - Aurora Health Center 84 South, Greenfield, Wisconsin
  - Aurora Surgery Centers LLC, Greenfield, Wisconsin
  - Aurora Medical Center Kenosha, Kenosha, Wisconsin
  - Mayo Clinic Health System- La Crosse, La Crosse, Wisconsin
  - Spine and Neuro, Health and Wellness Center, LLC, Lake Geneva, Wisconsin
  - Madison Surgery Center, Madison, Wisconsin
  - SSM Health - St. Mary's Hospital, Madison, Wisconsin
  - Marshfield Clinic Health System, Marshfield, Wisconsin
  - Drexel Town Square Surg Ctr, Menomonee Falls, Wisconsin
  - Froedtert Integrated Svc, Menomonee Falls, Wisconsin
  - West Bend Surg Ctr, Menomonee Falls, Wisconsin
  - Mayo Clinic Health System, Menomonie, Wisconsin
  - Aurora St Lukes Med Ctr, Milwaukee, Wisconsin
  - Aurora St Lukes Medical Center, Milwaukee, Wisconsin
  - WI Surgery Center, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua, Minocqua, Wisconsin
  - Aurora Health Care Southern Lakes, Inc, Mount Pleasant, Wisconsin
  - Advance Spine Ctr of Wisconsin, Neenah, Wisconsin
  - ThedaCare Inc. - Neenah, Neenah, Wisconsin
  - Aurora Medical Center Oshkosh, Oshkosh, Wisconsin
  - Spine Solutions of Sheboygan, LLC, Sheboygan, Wisconsin
  - Wisconsin Spine and Pain Surg Ctr, Sheboygan, Wisconsin
  - Door County Memorial Hospital, Sturgeon Bay, Wisconsin
  - Aurora Health Care Southern Lakes, Inc., Waukesha, Wisconsin
  - Aurora Med Ctr, Wauwatosa, Wisconsin
  - Wauwatosa Surgery Center, Wauwatosa, Wisconsin
  - Spine Solutions of West Bend, West Bend, Wisconsin
  - Wisconsin Spine and Pain West Bend, West Bend, Wisconsin
  - Evanston Regional Hospital, Evanston, Wyoming
  - Mem Hosp of Carbon County, Rawlins, Wyoming

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Staats PS, Hagedorn JM, Reece DE, Strand NH, Poree L. Percutaneous image-guided lumbar decompression and interspinous spacers for the treatment of lumbar spinal stenosis: A 2-year Medicare Claims Benchmark Study. Pain Pract. 2023 Sep;23(7):776-784. doi: 10.1111/papr.13256. Epub 2023 May 30. PMID 37254613
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/37254613/